CLINICAL TRIAL: NCT00938587
Title: A PHASE 2A, RANDOMIZED, DOUBLE-BLIND, ACTIVE AND PLACEBO-CONTROLLED STUDY OF PF-04171327 IN THE TREATMENT OF THE SIGNS AND SYMPTOMS OF RHEUMATOID ARTHRITIS
Brief Title: A Study Of PF-04171327 In The Treatment Of The Signs And Symptoms Of Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A9391005; 2009-013223-37 (EudraCT Number)
Record Dates: First submitted 2009-07-13; First posted 2009-07-14 (Estimated); Results first posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis Glucocorticoids Prednisone
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — fosdagrocorat; Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- PF-04171327 10 mg (Experimental)
  Interventions: Drug: PF-04171327 10 mg; Other: Prednisone Placebo
- PF-04171327 25 mg (Experimental)
  Interventions: Drug: PF-04171327 25 mg; Other: Prednisone Placebo
- Prednisone (Active Comparator)
  Interventions: Drug: Prednisone 5 mg; Other: Placebo for PF-04171327
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo; Other: Placebo for PF-04171327

INTERVENTIONS:
Drug: PF-04171327 10 mg — PF-04171327 10 mg tablet every day for 14 days
  Arms: PF-04171327 10 mg
Other: Prednisone Placebo — Placebo for Prednisone 5 mg tablet every day for 14 days
  Arms: PF-04171327 10 mg
Drug: PF-04171327 25 mg — PF-04171327 25 mg tablet every day for 14 days
  Arms: PF-04171327 25 mg
Other: Prednisone Placebo — Placebo for Prednisone 5 mg tablet every day for 14 days
  Arms: PF-04171327 25 mg
Drug: Prednisone 5 mg — Prednisone 5 mg tablet every day for 14 days
  Arms: Prednisone
Other: Placebo for PF-04171327 — Placebo for PF-04171327 every day for 14 days
  Arms: Prednisone
Other: Placebo — Placebo tablet every day for 14 days
  Arms: Placebo
Other: Placebo for PF-04171327 — Placebo tablet every day for 14 days
  Arms: Placebo

SUMMARY:
This study will investigate the safety and efficacy of an investigational drug, PF-04171327 on the signs and symptoms of rheumatoid arthritis in patients that require glucocorticoids while on background methotrexate. This study will also look at the response of chemical and biological markers in rheumatoid arthritis patients. Lastly, this study will measure the PK (amount of drug in the blood) of methotrexate while patients may be taking PF-04171327.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age, diagnosed with rheumatoid arthritis for a minimum duration of 3 months
* On stable dose of methotrexate for at least 6 weeks prior to screening
* Patient must have minimum disease activity level of ≥ 6 tender/painful joints, ≥ 6 swollen joints and CRP ≥ 0.7 mg/dL
* Not currently receiving steroid medication

Exclusion Criteria:

* Pregnant or nursing women
* Patients that have active infections, TB, HIV and/or Hepatitis B or C
* Patients that have a history of intolerance or significant adverse effects with the use of glucocorticoids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2009-10-07 (Actual); Primary Completion 2010-07-29 (Actual); Study Completion 2010-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (41):
- United States (10):
  - Anniston Medical Clinic, PC, Anniston, Alabama
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - Allergy, Asthma, Arthritis and Lung, Daytona Beach, Florida
  - Elite Research Institute, Miami, Florida
  - Millennium Research, Ormond Beach, Florida
  - Florida Medical Clinic, PA, Zephyrhills, Florida
  - The Arthritis Center, Springfield, Illinois
  - Premier Imaging Center, Bingham Farms, Michigan
  - Quest Research Institute, Bingham Farms, Michigan
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
- Czechia (5):
  - MEDIPONT Plus, s.r.o., České Budějovice
  - ARTMEDI UPD s r.o., Hostivice
  - Revmatologicka ambulance, Prague
  - Fakultni Thomayerova nemocnice s poliklinikou, Prague
  - DC Mediscan, Praha 11 - Chodov
- Centre for Assessment and Treatment of Rheumatic Diseases, Department of Medicine and Geriatrics, New Territories, Hong Kong
- Hungary (4):
  - Dr. Rethy Pal Korhaz es Rendelointezet\Reumatologia, Békéscsaba
  - Synexus Magyarorszag Kft., Budapest
  - Debreceni Egyetem Orvos és Egeszsegtudomanyi Centrum, Debrecen
  - MAV Korhaz es Rendelointezet, Szolnok
- Russia (4):
  - Moscow SHI City Clinical Hospital #4, Department of Therapy of Moscow Faculty, Moscow
  - Institution of Russian Academy of Medical Sciences Research Institute of Rheumatology RAMS, Moscow
  - SI Saint-Petersburg SRI for Emergency Care named after I.I. Dzhanelidze, Saint Petersburg
  - Regional State Institution of Healthcare Smolensk Regional Clinical Hospital, Smolensk
- Serbia (2):
  - Institute of Rheumatology, Belgrade
  - Institute for Rheumatic and Cardiovascular Disease Niska Banja, Niška Banja
- Changi General Hospital, Singapore, Singapore
- Slovakia (2):
  - Narodny ustav reumatickych chorob, Klinicke oddelenie, Piešťany
  - Nestatna reumatologicka ambulancia, MUDr. Pavol Polak, s.r.o., Žilina
- Severance Hospital, Yonsei University College of Medicine, Rheumatology, Internal Medicine, Seoul, South Korea
- Spain (4):
  - Hospital Nuestra Señora de La Esperanza, Santiago de Compostela, A Coruña
  - Hospital de Cruces, Barakaldo, Bilbao
  - Hospital de Basurto, Bilbao, Vizcaya
  - Hospital Universitario Virgen Macarena, Seville
- Taichung Veterans General Hospital, Taichung, Taiwan
- Ankara University School fo Medicine, Ankara, Turkey (Türkiye)
- Ukraine (5):
  - Chair of Cardiology & Functional Diagnostic, Kharkiv
  - State Institution "Institute of Gerontology of AMS of Ukraine", Kyiv
  - State Institution 'Institute of Gerontology of AMS of Ukraine', Kyiv
  - Municipal City Clinical Hospital #4, Department of Rheumatology, Lviv
  - Vinnitsa Regional Clinical Hospital n.a. Pirogov, Vinnitsa

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9391005&StudyName=A%20Study%20Of%20PF-04171327%20In%20The%20Treatment%20Of%20The%20Signs%20And%20Symptoms%20Of%20Rheumatoid%20Arthritis

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-04171327 10 mg + Placebo: Participants with rheumatoid arthritis (RA) received single oral dose of PF-04171327 10 milligram (mg) tablet and placebo matched to prednisone 5 mg capsule, once daily from Day 1 to Day 14. Participants were followed up to 31 days after last dose of study medication.
- PF-04171327 25 mg + Placebo: Participants with RA received single oral dose of PF-04171327 25 mg tablet and placebo matched to prednisone 5 mg capsule, once daily from Day 1 to Day 14. Participants were followed up to 31 days after last dose of study medication.
- Prednisone 5 mg + Placebo: Participants with RA received single oral dose of prednisone 5 mg capsule and placebo matched to PF-04171327 tablet, once daily from Day 1 to Day 14. Participants were followed up to 31 days after last dose of study medication.
- Placebo: Participants with RA received single oral dose of placebo, matched to PF-04171327 tablet and prednisone capsule, once daily from Day 1 to Day 14. Participants were followed up to 31 days after last dose of study medication.
Period: Overall Study
Arm/Group | PF-04171327 10 mg + Placebo | PF-04171327 25 mg + Placebo | Prednisone 5 mg + Placebo | Placebo
Started | 21 | 22 | 21 | 22
Completed | 18 | 21 | 20 | 20
Not Completed | 3 | 1 | 1 | 2
Not completed — Adverse Event | 2 | 0 | 0 | 2
Not completed — Did not meet entrance criteria | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all randomized participants who received at least 1 dose of the randomized investigational drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-04171327 10 mg + Placebo | PF-04171327 25 mg + Placebo | Prednisone 5 mg + Placebo | Placebo | Total
Number analyzed (Participants) | 21 | 22 | 21 | 22 | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (12.2) | 55.6 (11.4) | 56.0 (8.4) | 53.8 (11.9) | 55.5 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 12 | 15 | 20 | 61
  Male | 7 | 10 | 6 | 2 | 25

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Disease Activity Score Based on 28-Joints Count and C-Reactive Protein (4 Variables) (DAS28-4 [CRP]) at Day 14
Description: DAS28-4 (CRP) examines progression or improvement of RA. It was assessed from swollen joint count (SJC) and tender joint count (TJC) using the 28 joints count, CRP (normal range of CRP is less than (<) 10 milligram per liter [mg/L], decrease in the level of CRP indicates reduction in inflammation) and participant global assessment (PGA) of disease activity (participant global assessment of diseases condition scores ranging from 0 [very well condition] to 100 [very poor condition], higher scores indicated greater affectation due to disease activity). Total DAS28-4 (CRP) transformed score range: 0 (least severe) to 10 (most severe), higher scores indicate more severe disease activity. DAS28-4 (CRP) scores: less than equal to (<=) 3.2 implied low disease activity; greater than (>) 3.2 to 5.1 implied moderate to high disease activity.
Time Frame: Baseline, Day 14
Population: The full analysis set (FAS) included all randomized participants who received at least 1 dose of the randomized investigational drug. Here, 'n' signifies those participants who were evaluable at specified time points, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-04171327 10 mg + Placebo | PF-04171327 25 mg + Placebo | Prednisone 5 mg + Placebo | Placebo
Number analyzed (Participants) | 21 | 22 | 21 | 22
units on a scale
  Baseline | 6.04 (0.869) | 6.14 (0.755) | 5.92 (0.658) | 6.03 (0.810)
  Change at Day 14: number analyzed (Participants) | 18 | 21 | 20 | 21
  Change at Day 14 | -1.79 (0.916) | -2.22 (1.307) | -1.15 (0.935) | -0.96 (0.970)
Statistical Analysis 1: Comparison: PF-04171327 10 mg + Placebo vs Placebo; Day 14: Treatment difference and its corresponding 90 percent (%) confidence interval (CI) was based on least squares (LS) mean difference using mixed-model repeated measure (MMRM) where treatment, time, treatment-by-time interaction were fixed effects, participant as random effect, baseline as the covariate and compound symmetry (CS) as covariance structure; Test type: Superiority or Other; p = 0.0141, MMRM; LS mean difference = -0.73, 90% CI 2-sided [-1.21 to -0.24], Standard Error of Mean 0.291
Statistical Analysis 2: Comparison: PF-04171327 25 mg + Placebo vs Placebo; Day 14: Treatment difference and its corresponding 90 % CI was based on LS mean difference using MMRM where treatment, time, treatment-by-time interaction were fixed effects, participant as random effect, baseline as the covariate and CS as covariance structure; Test type: Superiority or Other; p < 0.0001, MMRM; LS mean difference = -1.26, 90% CI 2-sided [-1.73 to -0.79], Standard Error of Mean 0.283

2. Secondary Outcome: Change From Baseline in Tender Joints Count at Day 7, 14, 42
Description: Number of tender joints was determined by examining 28 joints and identified the joints that were painful under pressure or to passive motion. The number of tender joints was recorded on the joint assessment form at each visit, no tenderness = 0, tenderness = 1.
Time Frame: Baseline, Day 7, 14, 42
Population: FAS included all randomized participants who received at least 1 dose of the randomized investigational drug. Here, 'n' signifies those participants who were evaluable at specified time points, respectively.
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | PF-04171327 10 mg + Placebo | PF-04171327 25 mg + Placebo | Prednisone 5 mg + Placebo | Placebo
Number analyzed (Participants) | 21 | 22 | 21 | 22
tender joints
  Baseline | 17.10 (6.670) | 16.86 (5.375) | 15.05 (4.489) | 17.09 (6.023)
  Change at Day 7: number analyzed (Participants) | 21 | 21 | 21 | 22
  Change at Day 7 | -5.14 (6.807) | -5.95 (5.617) | -3.05 (4.117) | -4.18 (4.584)
  Change at Day 14: number analyzed (Participants) | 18 | 21 | 20 | 21
  Change at Day 14 | -7.22 (6.367) | -8.14 (6.755) | -4.15 (7.569) | -5.67 (6.807)
  Change at Day 42: number analyzed (Participants) | 19 | 21 | 20 | 21
  Change at Day 42 | -5.21 (6.188) | -6.52 (6.743) | -5.10 (6.703) | -6.81 (5.733)
Statistical Analysis 1: Comparison: PF-04171327 10 mg + Placebo vs Prednisone 5 mg + Placebo; Day 7: Treatment difference and its corresponding 90% CI was based on LS mean difference using MMRM where treatment, time, treatment-by-time interaction were fixed effects, participant as random effect, baseline as the covariate and CS as covariance structure; Test type: Superiority or Other; p = 0.4370, MMRM; LS mean difference = -1.45, 90% CI 2-sided [-4.54 to 1.63], Standard Error of Mean 1.865
Statistical Analysis 2: Comparison: PF-04171327 25 mg + Placebo vs Prednisone 5 mg + Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.1802, MMRM; LS mean difference = -2.50, 90% CI 2-sided [-5.58 to 0.57], Standard Error of Mean 1.858
Statistical Analysis 3: Comparison: PF-04171327 10 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.6012, MMRM; LS mean difference = -0.96, 90% CI 2-sided [-3.99 to 2.07], Standard Error of Mean 1.832
Statistical Analysis 4: Comparison: PF-04171327 25 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.2753, MMRM; LS mean difference = -2.01, 90% CI 2-sided [-5.04 to 1.03], Standard Error of Mean 1.834
Statistical Analysis 5: Comparison: Prednisone 5 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.7892, MMRM; LS mean difference = 0.49, 90% CI 2-sided [-2.56 to 3.55], Standard Error of Mean 1.844
Statistical Analysis 6: Comparison: PF-04171327 10 mg + Placebo vs Prednisone 5 mg + Placebo; Day 14: Treatment difference and its corresponding 90% CI was based on LS mean difference using MMRM where treatment, time, treatment-by-time interaction were fixed effects, participant as random effect, baseline as the covariate and CS as covariance structure; Test type: Superiority or Other; p = 0.3765, MMRM; LS mean difference = -1.72, 90% CI 2-sided [-4.92 to 1.49], Standard Error of Mean 1.937
Statistical Analysis 7: Comparison: PF-04171327 25 mg + Placebo vs Prednisone 5 mg + Placebo; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.0571, MMRM; LS mean difference = -3.59, 90% CI 2-sided [-6.69 to -0.49], Standard Error of Mean 1.873
Statistical Analysis 8: Comparison: PF-04171327 10 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.6553, MMRM; LS mean difference = -0.85, 90% CI 2-sided [-3.99 to 2.29], Standard Error of Mean 1.896
Statistical Analysis 9: Comparison: PF-04171327 25 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.1427, MMRM; LS mean difference = -2.72, 90% CI 2-sided [-5.78 to 0.33], Standard Error of Mean 1.847
Statistical Analysis 10: Comparison: Prednisone 5 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.6430, MMRM; LS mean difference = 0.87, 90% CI 2-sided [-2.23 to 3.97], Standard Error of Mean 1.873
Statistical Analysis 11: Comparison: PF-04171327 10 mg + Placebo vs Prednisone 5 mg + Placebo; Day 42: Treatment difference and its corresponding 90% CI was based on LS mean difference using MMRM where treatment, time, treatment-by-time interaction were fixed effects, participant as random effect, baseline as the covariate and CS as covariance structure; Test type: Superiority or Other; p = 0.5868, MMRM; LS mean difference = 1.04, 90% CI 2-sided [-2.13 to 4.22], Standard Error of Mean 1.918
Statistical Analysis 12: Comparison: PF-04171327 25 mg + Placebo vs Prednisone 5 mg + Placebo; [analysis description as in outcome 2, analysis 11]; Test type: Superiority or Other; p = 0.5860, MMRM; LS mean difference = -1.02, 90% CI 2-sided [-4.12 to 2.08], Standard Error of Mean 1.873
Statistical Analysis 13: Comparison: PF-04171327 10 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 11]; Test type: Superiority or Other; p = 0.3288, MMRM; LS mean difference = 1.84, 90% CI 2-sided [-1.27 to 4.95], Standard Error of Mean 1.879
Statistical Analysis 14: Comparison: PF-04171327 25 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 11]; Test type: Superiority or Other; p = 0.9027, MMRM; LS mean difference = -0.23, 90% CI 2-sided [-3.28 to 2.83], Standard Error of Mean 1.846
Statistical Analysis 15: Comparison: Prednisone 5 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 11]; Test type: Superiority or Other; p = 0.6710, MMRM; LS mean difference = 0.80, 90% CI 2-sided [-2.30 to 3.89], Standard Error of Mean 1.871

3. Secondary Outcome: Change From Baseline in Swollen Joints Count at Day 7, 14 and 42
Description: Number of swollen joints was determined by examination of 28 joints and identifying if swelling was present. The number of swollen joints was recorded on the joint assessment form at each visit, no swelling = 0, swelling =1.
Time Frame: Baseline, Day 7, 14, 42
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | PF-04171327 10 mg + Placebo | PF-04171327 25 mg + Placebo | Prednisone 5 mg + Placebo | Placebo
Number analyzed (Participants) | 21 | 22 | 21 | 22
swollen joints
  Baseline | 11.95 (4.717) | 11.73 (4.038) | 10.67 (3.554) | 11.64 (4.065)
  Change at Day 7: number analyzed (Participants) | 21 | 21 | 21 | 22
  Change at Day 7 | -3.19 (3.544) | -5.19 (4.045) | -2.90 (3.048) | -2.91 (3.963)
  Change at Day 14: number analyzed (Participants) | 18 | 21 | 20 | 21
  Change at Day 14 | -5.50 (3.777) | -6.71 (4.256) | -4.85 (3.133) | -5.24 (4.816)
  Change at Day 42: number analyzed (Participants) | 19 | 21 | 20 | 21
  Change at Day 42 | -3.26 (3.679) | -4.81 (4.167) | -6.15 (3.787) | -4.71 (4.900)
Statistical Analysis 1: Comparison: PF-04171327 10 mg + Placebo vs Prednisone 5 mg + Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.8370, MMRM; LS mean difference = 0.23, 90% CI 2-sided [-1.63 to 2.09], Standard Error of Mean 1.123
Statistical Analysis 2: Comparison: PF-04171327 25 mg + Placebo vs Prednisone 5 mg + Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0819, MMRM; LS mean difference = -1.96, 90% CI 2-sided [-3.81 to -0.11], Standard Error of Mean 1.120
Statistical Analysis 3: Comparison: PF-04171327 10 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.8892, MMRM; LS mean difference = -0.15, 90% CI 2-sided [-1.98 to 1.67], Standard Error of Mean 1.106
Statistical Analysis 4: Comparison: PF-04171327 25 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0353, MMRM; LS mean difference = -2.35, 90% CI 2-sided [-4.17 to -0.52], Standard Error of Mean 1.106
Statistical Analysis 5: Comparison: Prednisone 5 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.7283, MMRM; LS mean difference = -0.39, 90% CI 2-sided [-2.22 to 1.45], Standard Error of Mean 1.108
Statistical Analysis 6: Comparison: PF-04171327 10 mg + Placebo vs Prednisone 5 mg + Placebo; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.9083, MMRM; LS mean difference = 0.14, 90% CI 2-sided [-1.81 to 2.08], Standard Error of Mean 1.174
Statistical Analysis 7: Comparison: PF-04171327 25 mg + Placebo vs Prednisone 5 mg + Placebo; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.1641, MMRM; LS mean difference = -1.58, 90% CI 2-sided [-3.45 to 0.29], Standard Error of Mean 1.132
Statistical Analysis 8: Comparison: PF-04171327 10 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.8170, MMRM; LS mean difference = 0.27, 90% CI 2-sided [-1.64 to 2.18], Standard Error of Mean 1.155
Statistical Analysis 9: Comparison: PF-04171327 25 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.1958, MMRM; LS mean difference = -1.45, 90% CI 2-sided [-3.29 to 0.40], Standard Error of Mean 1.116
Statistical Analysis 10: Comparison: Prednisone 5 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.9070, MMRM; LS mean difference = 0.13, 90% CI 2-sided [-1.74 to 2.00], Standard Error of Mean 1.130
Statistical Analysis 11: Comparison: PF-04171327 10 mg + Placebo vs Prednisone 5 mg + Placebo; [analysis description as in outcome 2, analysis 11]; Test type: Superiority or Other; p = 0.0023, MMRM; LS mean difference = 3.58, 90% CI 2-sided [1.67 to 5.50], Standard Error of Mean 1.160
Statistical Analysis 12: Comparison: PF-04171327 25 mg + Placebo vs Prednisone 5 mg + Placebo; [analysis description as in outcome 2, analysis 11]; Test type: Superiority or Other; p = 0.1531, MMRM; LS mean difference = 1.62, 90% CI 2-sided [-0.25 to 3.49], Standard Error of Mean 1.132
Statistical Analysis 13: Comparison: PF-04171327 10 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 11]; Test type: Superiority or Other; p = 0.1506, MMRM; LS mean difference = 1.65, 90% CI 2-sided [-0.24 to 3.53], Standard Error of Mean 1.141
Statistical Analysis 14: Comparison: PF-04171327 25 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 11]; Test type: Superiority or Other; p = 0.7800, MMRM; LS mean difference = -0.31, 90% CI 2-sided [-2.16 to 1.53], Standard Error of Mean 1.116
Statistical Analysis 15: Comparison: Prednisone 5 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 11]; Test type: Superiority or Other; p = 0.0883, MMRM; LS mean difference = -1.94, 90% CI 2-sided [-3.80 to -0.07], Standard Error of Mean 1.130

4. Secondary Outcome: Change From Baseline in C-Reactive Protein (CRP) at Day 7, 14 and 42
Description: The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. Normal range of CRP is less than (<) 10 mg/L. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement.
Time Frame: Baseline, Day 7, 14, 42
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | PF-04171327 10 mg + Placebo | PF-04171327 25 mg + Placebo | Prednisone 5 mg + Placebo | Placebo
Number analyzed (Participants) | 21 | 22 | 21 | 22
mg/L
  Baseline | 20.24 (16.431) | 30.15 (35.396) | 20.02 (14.022) | 16.97 (19.580)
  Change at Day 7: number analyzed (Participants) | 20 | 21 | 21 | 21
  Change at Day 7 | -13.78 (18.208) | -23.60 (32.808) | -4.64 (18.487) | 1.31 (16.374)
  Change at Day 14: number analyzed (Participants) | 18 | 21 | 20 | 21
  Change at Day 14 | -18.13 (17.519) | -24.12 (33.273) | -7.63 (16.876) | -1.32 (10.357)
  Change at Day 42: number analyzed (Participants) | 19 | 21 | 20 | 21
  Change at Day 42 | 3.14 (28.198) | -13.09 (27.448) | -8.02 (13.850) | -5.11 (23.304)
Statistical Analysis 1: Comparison: PF-04171327 10 mg + Placebo vs Prednisone 5 mg + Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0599, MMRM; LS mean difference = -8.47, 90% CI 2-sided [-15.87 to -1.07], Standard Error of Mean 4.480
Statistical Analysis 2: Comparison: PF-04171327 25 mg + Placebo vs Prednisone 5 mg + Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0030, MMRM; LS mean difference = -13.29, 90% CI 2-sided [-20.61 to -5.96], Standard Error of Mean 4.436
Statistical Analysis 3: Comparison: PF-04171327 10 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0053, MMRM; LS mean difference = -12.63, 90% CI 2-sided [-20.03 to -5.22], Standard Error of Mean 4.483
Statistical Analysis 4: Comparison: PF-04171327 25 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0001, MMRM; LS mean difference = -17.44, 90% CI 2-sided [-24.78 to -10.10], Standard Error of Mean 4.445
Statistical Analysis 5: Comparison: Prednisone 5 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.3492, MMRM; LS mean difference = -4.15, 90% CI 2-sided [-11.46 to 3.16], Standard Error of Mean 4.427
Statistical Analysis 6: Comparison: PF-04171327 10 mg + Placebo vs Prednisone 5 mg + Placebo; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.0389, MMRM; LS mean difference = -9.68, 90% CI 2-sided [-17.38 to -1.98], Standard Error of Mean 4.661
Statistical Analysis 7: Comparison: PF-04171327 25 mg + Placebo vs Prednisone 5 mg + Placebo; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.0142, MMRM; LS mean difference = -11.10, 90% CI 2-sided [-18.51 to -3.68], Standard Error of Mean 4.490
Statistical Analysis 8: Comparison: PF-04171327 10 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.0037, MMRM; LS mean difference = -13.51, 90% CI 2-sided [-21.13 to -5.89], Standard Error of Mean 4.612
Statistical Analysis 9: Comparison: PF-04171327 25 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.0009, MMRM; LS mean difference = -14.93, 90% CI 2-sided [-22.27 to -7.58], Standard Error of Mean 4.447
Statistical Analysis 10: Comparison: Prednisone 5 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.3939, MMRM; LS mean difference = -3.83, 90% CI 2-sided [-11.23 to 3.57], Standard Error of Mean 4.484
Statistical Analysis 11: Comparison: PF-04171327 10 mg + Placebo vs Prednisone 5 mg + Placebo; [analysis description as in outcome 2, analysis 11]; Test type: Superiority or Other; p = 0.0127, MMRM; LS mean difference = 11.54, 90% CI 2-sided [3.95 to 19.13], Standard Error of Mean 4.595
Statistical Analysis 12: Comparison: PF-04171327 25 mg + Placebo vs Prednisone 5 mg + Placebo; [analysis description as in outcome 2, analysis 11]; Test type: Superiority or Other; p = 0.9425, MMRM; LS mean difference = 0.32, 90% CI 2-sided [-7.09 to 7.74], Standard Error of Mean 4.490
Statistical Analysis 13: Comparison: PF-04171327 10 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 11]; Test type: Superiority or Other; p = 0.0155, MMRM; LS mean difference = 11.08, 90% CI 2-sided [3.58 to 18.59], Standard Error of Mean 4.544
Statistical Analysis 14: Comparison: PF-04171327 25 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 11]; Test type: Superiority or Other; p = 0.9757, MMRM; LS mean difference = -0.14, 90% CI 2-sided [-7.48 to 7.21], Standard Error of Mean 4.447
Statistical Analysis 15: Comparison: Prednisone 5 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 11]; Test type: Superiority or Other; p = 0.9184, MMRM; LS mean difference = -0.46, 90% CI 2-sided [-7.86 to 6.94], Standard Error of Mean 4.484

5. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) Score at Day 7 and 14
Description: HAQ-DI assessed the ability of participants to perform task in 8 domains of daily living activities: dress/groom, arise, eat, walk, reach, grip, hygiene, and common activities. Each item was scored on a 4-point scale ranging from 0 to 3: 0= no difficulty; 1= some difficulty; 2= much difficulty; 3= unable to do, higher scores indicate more difficulty. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible HAQ-DI score range: 0 (no difficulty) to 3 (extreme difficulty), where higher scores indicate more difficulty while performing daily living activities.
Time Frame: Baseline, Day 7, 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-04171327 10 mg + Placebo | PF-04171327 25 mg + Placebo | Prednisone 5 mg + Placebo | Placebo
Number analyzed (Participants) | 21 | 22 | 21 | 22
units on a scale
  Baseline | 1.76 (0.831) | 1.41 (0.796) | 1.62 (0.498) | 1.73 (0.935)
  Change at Day 7: number analyzed (Participants) | 21 | 21 | 21 | 21
  Change at Day 7 | -0.24 (0.700) | -0.24 (0.700) | -0.24 (0.436) | -0.10 (0.539)
  Change at Day 14: number analyzed (Participants) | 19 | 21 | 20 | 21
  Change at Day 14 | -0.58 (1.017) | -0.43 (0.870) | -0.25 (0.550) | -0.24 (0.768)
Statistical Analysis 1: Comparison: PF-04171327 10 mg + Placebo vs Prednisone 5 mg + Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.2403, MMRM; LS mean difference = -0.16, 90% CI 2-sided [-0.38 to 0.06], Standard Error of Mean 0.135
Statistical Analysis 2: Comparison: PF-04171327 25 mg + Placebo vs Prednisone 5 mg + Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0270, MMRM; LS mean difference = -0.30, 90% CI 2-sided [-0.52 to -0.08], Standard Error of Mean 0.134
Statistical Analysis 3: Comparison: PF-04171327 10 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.3139, MMRM; LS mean difference = -0.13, 90% CI 2-sided [-0.36 to 0.09], Standard Error of Mean 0.133
Statistical Analysis 4: Comparison: PF-04171327 25 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0415, MMRM; LS mean difference = -0.28, 90% CI 2-sided [-0.50 to -0.05], Standard Error of Mean 0.134
Statistical Analysis 5: Comparison: Prednisone 5 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.8585, MMRM; LS mean difference = 0.02, 90% CI 2-sided [-0.20 to 0.25], Standard Error of Mean 0.134
Statistical Analysis 6: Comparison: PF-04171327 10 mg + Placebo vs Prednisone 5 mg + Placebo; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.7284, MMRM; LS mean difference = -0.05, 90% CI 2-sided [-0.28 to 0.18], Standard Error of Mean 0.138
Statistical Analysis 7: Comparison: PF-04171327 25 mg + Placebo vs Prednisone 5 mg + Placebo; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.0171, MMRM; LS mean difference = -0.33, 90% CI 2-sided [-0.55 to -0.10], Standard Error of Mean 0.135
Statistical Analysis 8: Comparison: PF-04171327 10 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.2277, MMRM; LS mean difference = -0.16, 90% CI 2-sided [-0.39 to 0.06], Standard Error of Mean 0.135
Statistical Analysis 9: Comparison: PF-04171327 25 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.0013, MMRM; LS mean difference = -0.44, 90% CI 2-sided [-0.67 to -0.22], Standard Error of Mean 0.134
Statistical Analysis 10: Comparison: Prednisone 5 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.3908, MMRM; LS mean difference = -0.12, 90% CI 2-sided [-0.34 to 0.11], Standard Error of Mean 0.135

6. Secondary Outcome: Change From Baseline in Participant Assessment of Arthritis Pain at Day 7 and 14
Description: Participant assessment of arthritis pain included assessment of severity of arthritis pain using a 100 millimeter (mm) visual analog scale (VAS). Participants placed a mark on the VAS between 0 mm (no pain) and 100 mm (most severe pain), which corresponded to the magnitude of their pain, higher scores indicate more pain.
Time Frame: Baseline, Day 7, 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | PF-04171327 10 mg + Placebo | PF-04171327 25 mg + Placebo | Prednisone 5 mg + Placebo | Placebo
Number analyzed (Participants) | 21 | 22 | 21 | 22
mm
  Baseline | 62.45 (25.586) | 60.49 (21.123) | 63.17 (15.551) | 66.65 (15.368)
  Change at Day 7: number analyzed (Participants) | 21 | 21 | 21 | 22
  Change at Day 7 | -12.03 (23.584) | -16.95 (25.056) | -8.67 (18.343) | -11.00 (21.889)
  Change at Day 14: number analyzed (Participants) | 19 | 21 | 20 | 21
  Change at Day 14 | -25.83 (31.899) | -27.29 (25.823) | -21.47 (23.627) | -14.69 (23.718)
Statistical Analysis 1: Comparison: PF-04171327 10 mg + Placebo vs Prednisone 5 mg + Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.6067, MMRM; LS mean difference = -3.66, 90% CI 2-sided [-15.43 to 8.10], Standard Error of Mean 7.093
Statistical Analysis 2: Comparison: PF-04171327 25 mg + Placebo vs Prednisone 5 mg + Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.1816, MMRM; LS mean difference = -9.55, 90% CI 2-sided [-21.32 to 2.23], Standard Error of Mean 7.101
Statistical Analysis 3: Comparison: PF-04171327 10 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.6873, MMRM; LS mean difference = -2.84, 90% CI 2-sided [-14.50 to 8.82], Standard Error of Mean 7.029
Statistical Analysis 4: Comparison: PF-04171327 25 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.2188, MMRM; LS mean difference = -8.72, 90% CI 2-sided [-20.42 to 2.98], Standard Error of Mean 7.052
Statistical Analysis 5: Comparison: Prednisone 5 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.9067, MMRM; LS mean difference = 0.83, 90% CI 2-sided [-10.82 to 12.47], Standard Error of Mean 7.024
Statistical Analysis 6: Comparison: PF-04171327 10 mg + Placebo vs Prednisone 5 mg + Placebo; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.5803, MMRM; LS mean difference = -4.02, 90% CI 2-sided [-16.05 to 8.00], Standard Error of Mean 7.254
Statistical Analysis 7: Comparison: PF-04171327 25 mg + Placebo vs Prednisone 5 mg + Placebo; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.2490, MMRM; LS mean difference = -8.29, 90% CI 2-sided [-20.16 to 3.57], Standard Error of Mean 7.156
Statistical Analysis 8: Comparison: PF-04171327 10 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.1081, MMRM; LS mean difference = -11.62, 90% CI 2-sided [-23.52 to 0.28], Standard Error of Mean 7.178
Statistical Analysis 9: Comparison: PF-04171327 25 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.0271, MMRM; LS mean difference = -15.89, 90% CI 2-sided [-27.66 to -4.12], Standard Error of Mean 7.098
Statistical Analysis 10: Comparison: Prednisone 5 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.2881, MMRM; LS mean difference = -7.60, 90% CI 2-sided [-19.41 to 4.21], Standard Error of Mean 7.121

7. Secondary Outcome: Change From Baseline in Participant Global Assessment (PGA) of Arthritis at Day 7 and 14
Description: PGA was a questionnaire where participants answered the following question, "Considering all the ways your arthritis affects you, how are you feeling today?" The participants' response were recorded using a 100 mm visual analog scale placing a mark on the scale, between 0 mm (very well condition) to 100 mm (very poor condition). Higher scores indicate higher degree of arthritis.
Time Frame: Baseline, Day 7, 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | PF-04171327 10 mg + Placebo | PF-04171327 25 mg + Placebo | Prednisone 5 mg + Placebo | Placebo
Number analyzed (Participants) | 21 | 22 | 21 | 22
mm
  Baseline | 60.71 (24.265) | 63.55 (20.589) | 65.89 (14.957) | 65.26 (18.426)
  Change at Day 7: number analyzed (Participants) | 21 | 21 | 21 | 22
  Change at Day 7 | -16.05 (21.800) | -18.75 (25.933) | -11.87 (17.036) | -7.94 (21.281)
  Change at Day 14: number analyzed (Participants) | 19 | 21 | 20 | 21
  Change at Day 14 | -22.63 (30.656) | -27.97 (26.894) | -22.43 (22.303) | -11.77 (27.457)
Statistical Analysis 1: Comparison: PF-04171327 10 mg + Placebo vs Prednisone 5 mg + Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.3579, MMRM; LS mean difference = -6.52, 90% CI 2-sided [-18.23 to 5.19], Standard Error of Mean 7.059
Statistical Analysis 2: Comparison: PF-04171327 25 mg + Placebo vs Prednisone 5 mg + Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.2274, MMRM; LS mean difference = -8.55, 90% CI 2-sided [-20.24 to 3.14], Standard Error of Mean 7.046
Statistical Analysis 3: Comparison: PF-04171327 10 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.1482, MMRM; LS mean difference = -10.15, 90% CI 2-sided [-21.72 to 1.41], Standard Error of Mean 6.973
Statistical Analysis 4: Comparison: PF-04171327 25 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0828, MMRM; LS mean difference = -12.19, 90% CI 2-sided [-23.74 to -0.64], Standard Error of Mean 6.962
Statistical Analysis 5: Comparison: Prednisone 5 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.6021, MMRM; LS mean difference = -3.64, 90% CI 2-sided [-15.17 to 7.90], Standard Error of Mean 6.953
Statistical Analysis 6: Comparison: PF-04171327 10 mg + Placebo vs Prednisone 5 mg + Placebo; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.7528, MMRM; LS mean difference = -2.28, 90% CI 2-sided [-14.24 to 9.68], Standard Error of Mean 7.213
Statistical Analysis 7: Comparison: PF-04171327 25 mg + Placebo vs Prednisone 5 mg + Placebo; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.2523, MMRM; LS mean difference = -8.17, 90% CI 2-sided [-19.94 to 3.60], Standard Error of Mean 7.100
Statistical Analysis 8: Comparison: PF-04171327 10 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.1049, MMRM; LS mean difference = -11.63, 90% CI 2-sided [-23.43 to 0.17], Standard Error of Mean 7.118
Statistical Analysis 9: Comparison: PF-04171327 25 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.0138, MMRM; LS mean difference = -17.53, 90% CI 2-sided [-29.14 to -5.91], Standard Error of Mean 7.006
Statistical Analysis 10: Comparison: Prednisone 5 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.1873, MMRM; LS mean difference = -9.36, 90% CI 2-sided [-21.05 to 2.34], Standard Error of Mean 7.052

8. Secondary Outcome: Change From Baseline in Physician Global Assessment (PhGA) of Arthritis at Day 7 and 14
Description: PhGA included assessment of severity of arthritis pain where physicians were asked to rate the severity of the participant's overall arthritis. The physician's response was recorded using a visual analog scale between 0 mm (very good condition) to 100 mm (very poor condition). Higher scores indicate higher degree of arthritis.
Time Frame: Baseline, Day 7, 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | PF-04171327 10 mg + Placebo | PF-04171327 25 mg + Placebo | Prednisone 5 mg + Placebo | Placebo
Number analyzed (Participants) | 21 | 22 | 21 | 22
mm
  Baseline | 58.10 (19.917) | 62.27 (13.016) | 57.86 (13.309) | 59.87 (15.194)
  Change at Day 7: number analyzed (Participants) | 21 | 21 | 21 | 22
  Change at Day 7 | -13.38 (22.295) | -20.42 (16.487) | -9.71 (13.723) | -13.58 (16.208)
  Change at Day 14: number analyzed (Participants) | 19 | 21 | 20 | 21
  Change at Day 14 | -22.16 (23.176) | -32.19 (19.473) | -20.90 (18.671) | -14.87 (21.176)
Statistical Analysis 1: Comparison: PF-04171327 10 mg + Placebo vs Prednisone 5 mg + Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.5090, MMRM; LS mean difference = -3.54, 90% CI 2-sided [-12.40 to 5.32], Standard Error of Mean 5.339
Statistical Analysis 2: Comparison: PF-04171327 25 mg + Placebo vs Prednisone 5 mg + Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0998, MMRM; LS mean difference = -8.89, 90% CI 2-sided [-17.78 to -0.01], Standard Error of Mean 5.354
Statistical Analysis 3: Comparison: PF-04171327 10 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.8866, MMRM; LS mean difference = -0.76, 90% CI 2-sided [-9.52 to 8.01], Standard Error of Mean 5.282
Statistical Analysis 4: Comparison: PF-04171327 25 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.2499, MMRM; LS mean difference = -6.11, 90% CI 2-sided [-14.88 to 2.66], Standard Error of Mean 5.280
Statistical Analysis 5: Comparison: Prednisone 5 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.5995, MMRM; LS mean difference = 2.78, 90% CI 2-sided [-5.99 to 11.55], Standard Error of Mean 5.283
Statistical Analysis 6: Comparison: PF-04171327 10 mg + Placebo vs Prednisone 5 mg + Placebo; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.9117, MMRM; LS mean difference = 0.60, 90% CI 2-sided [-8.40 to 9.61], Standard Error of Mean 5.429
Statistical Analysis 7: Comparison: PF-04171327 25 mg + Placebo vs Prednisone 5 mg + Placebo; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.0684, MMRM; LS mean difference = -9.91, 90% CI 2-sided [-18.84 to -0.98], Standard Error of Mean 5.381
Statistical Analysis 8: Comparison: PF-04171327 10 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.2292, MMRM; LS mean difference = -6.49, 90% CI 2-sided [-15.39 to 2.42], Standard Error of Mean 5.366
Statistical Analysis 9: Comparison: PF-04171327 25 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.0018, MMRM; LS mean difference = -17.00, 90% CI 2-sided [-25.81 to -8.19], Standard Error of Mean 5.308
Statistical Analysis 10: Comparison: Prednisone 5 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.1867, MMRM; LS mean difference = -7.09, 90% CI 2-sided [-15.95 to 1.76], Standard Error of Mean 5.337

9. Secondary Outcome: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) Version 2.0 (V2) at Day 14
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and well-being: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional and mental health. Score for each of the 8 aspects are scaled from 0 (worst condition) to 100 (best condition), where higher scores indicate better health status. These 8 domains were also reported as two summary scores: physical component scores and mental component scores. Score range for each of the 2 summary scores = 0 (worst condition) to 100 (best condition), where higher scores represent better health status.
Time Frame: Baseline, Day 14 (D14)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-04171327 10 mg + Placebo | PF-04171327 25 mg + Placebo | Prednisone 5 mg + Placebo | Placebo
Number analyzed (Participants) | 21 | 22 | 21 | 22
units on a scale
  Baseline: Physical functioning | 29.92 (9.624) | 30.69 (8.305) | 29.14 (7.187) | 32.74 (9.904)
  Change at D14: Physical functioning: number analyzed (Participants) | 19 | 21 | 20 | 20
  Change at D14: Physical functioning | 4.52 (9.142) | 4.58 (6.660) | 4.71 (6.543) | 0.51 (10.968)
  Baseline: Role physical | 35.72 (9.452) | 35.69 (8.680) | 33.10 (7.288) | 34.28 (10.031)
  Change at D14: Role physical: number analyzed (Participants) | 19 | 21 | 20 | 20
  Change at D14: Role physical | 4.27 (12.182) | 7.27 (9.378) | 5.01 (6.789) | 5.97 (10.516)
  Baseline: Bodily pain | 31.41 (7.473) | 32.88 (6.234) | 31.35 (4.159) | 33.43 (6.851)
  Change at D14: Bodily pain: number analyzed (Participants) | 19 | 21 | 20 | 20
  Change at D14: Bodily pain | 11.25 (11.394) | 11.60 (7.609) | 7.73 (6.435) | 4.33 (11.369)
  Baseline: General health | 30.91 (9.564) | 37.33 (11.005) | 35.36 (8.423) | 35.43 (9.408)
  Change at D14: General health: number analyzed (Participants) | 19 | 21 | 20 | 20
  Change at D14: General health | 4.40 (6.604) | 3.96 (5.853) | 3.31 (5.652) | 4.09 (6.740)
  Baseline: Vitality | 38.98 (10.166) | 42.43 (9.891) | 39.70 (8.671) | 39.98 (8.567)
  Change at D14: Vitality: number analyzed (Participants) | 19 | 21 | 20 | 20
  Change at D14: Vitality | 7.88 (11.603) | 7.70 (7.183) | 4.79 (7.229) | 4.19 (10.962)
  Baseline: Social functioning | 39.50 (10.384) | 39.05 (12.411) | 34.89 (9.468) | 35.87 (11.809)
  Change at D14: Social functioning: number analyzed (Participants) | 19 | 21 | 20 | 20
  Change at D14: Social functioning | 4.25 (10.988) | 7.68 (9.090) | 5.65 (5.647) | 4.57 (10.934)
  Baseline: Role emotional | 36.39 (13.164) | 37.95 (12.978) | 35.49 (12.287) | 35.37 (14.477)
  Change at D14: Role emotional: number analyzed (Participants) | 19 | 21 | 20 | 20
  Change at D14: Role emotional | 5.18 (15.873) | 6.31 (12.051) | 2.65 (12.888) | 2.65 (14.538)
  Baseline: Mental health | 37.71 (14.742) | 42.40 (11.681) | 37.97 (11.807) | 36.23 (12.871)
  Change at D14: Mental health: number analyzed (Participants) | 19 | 21 | 20 | 20
  Change at D14: Mental health | 7.00 (15.072) | 4.62 (9.368) | 5.13 (8.540) | 2.49 (11.819)
  Baseline: Physical component | 30.89 (7.342) | 32.05 (6.627) | 30.91 (5.185) | 33.93 (6.554)
  Change at D14: Physical component: number analyzed (Participants) | 19 | 21 | 20 | 20
  Change at D14: Physical component | 5.74 (6.611) | 7.10 (4.351) | 5.49 (5.219) | 3.73 (8.594)
  Baseline: Mental component | 41.19 (14.648) | 44.42 (13.036) | 40.30 (12.464) | 38.55 (13.064)
  Change at D14: Mental component: number analyzed (Participants) | 19 | 21 | 20 | 20
  Change at D14: Mental component | 5.91 (14.065) | 5.72 (9.743) | 3.78 (8.358) | 3.24 (12.812)
Statistical Analysis 1: Comparison: PF-04171327 10 mg + Placebo vs Prednisone 5 mg + Placebo; Physical functioning at D14: Treatment difference and its corresponding 90% CI was based on LS mean difference using analysis of covariance (ANCOVA) where treatment as fixed effect, baseline as the covariate; Test type: Superiority or Other; p = 0.9624, ANCOVA; LS mean difference = -0.13, 90% CI 2-sided [-4.64 to 4.38], Standard Error of Mean 2.708
Statistical Analysis 2: Comparison: PF-04171327 25 mg + Placebo vs Prednisone 5 mg + Placebo; Physical functioning at D14: Treatment difference and its corresponding 90% CI was based on LS mean difference using ANCOVA where treatment as fixed effect, baseline as the covariate; Test type: Superiority or Other; p = 0.9493, ANCOVA; LS mean difference = 0.17, 90% CI 2-sided [-4.24 to 4.58], Standard Error of Mean 2.650
Statistical Analysis 3: Comparison: PF-04171327 10 mg + Placebo vs Placebo; [analysis description as in outcome 9, analysis 2]; Test type: Superiority or Other; p = 0.2100, ANCOVA; LS mean difference = 3.46, 90% CI 2-sided [-1.10 to 8.02], Standard Error of Mean 2.738
Statistical Analysis 4: Comparison: PF-04171327 25 mg + Placebo vs Placebo; [analysis description as in outcome 9, analysis 2]; Test type: Superiority or Other; p = 0.1602, ANCOVA; LS mean difference = 3.76, 90% CI 2-sided [-0.66 to 8.18], Standard Error of Mean 2.651
Statistical Analysis 5: Comparison: Prednisone 5 mg + Placebo vs Placebo; [analysis description as in outcome 9, analysis 2]; Test type: Superiority or Other; p = 0.1892, ANCOVA; LS mean difference = 3.59, 90% CI 2-sided [-0.92 to 8.10], Standard Error of Mean 2.710
Statistical Analysis 6: Comparison: PF-04171327 10 mg + Placebo vs Prednisone 5 mg + Placebo; Role physical at D14: Treatment difference and its corresponding 90% CI was based on LS mean difference using ANCOVA where treatment as fixed effect, baseline as the covariate; Test type: Superiority or Other; p = 0.7899, ANCOVA; LS mean difference = 0.74, 90% CI 2-sided [-3.89 to 5.38], Standard Error of Mean 2.781
Statistical Analysis 7: Comparison: PF-04171327 25 mg + Placebo vs Prednisone 5 mg + Placebo; [analysis description as in outcome 9, analysis 6]; Test type: Superiority or Other; p = 0.1490, ANCOVA; LS mean difference = 3.96, 90% CI 2-sided [-0.56 to 8.49], Standard Error of Mean 2.719
Statistical Analysis 8: Comparison: PF-04171327 10 mg + Placebo vs Placebo; [analysis description as in outcome 9, analysis 6]; Test type: Superiority or Other; p = 0.6238, ANCOVA; LS mean difference = -1.36, 90% CI 2-sided [-5.97 to 3.24], Standard Error of Mean 2.766
Statistical Analysis 9: Comparison: PF-04171327 25 mg + Placebo vs Placebo; [analysis description as in outcome 9, analysis 6]; Test type: Superiority or Other; p = 0.4933, ANCOVA; LS mean difference = 1.86, 90% CI 2-sided [-2.64 to 6.35], Standard Error of Mean 2.699
Statistical Analysis 10: Comparison: Prednisone 5 mg + Placebo vs Placebo; [analysis description as in outcome 9, analysis 6]; Test type: Superiority or Other; p = 0.4445, ANCOVA; LS mean difference = -2.11, 90% CI 2-sided [-6.67 to 2.46], Standard Error of Mean 2.739
Statistical Analysis 11: Comparison: PF-04171327 10 mg + Placebo vs Prednisone 5 mg + Placebo; Bodily pain at D14: Treatment difference and its corresponding 90% CI was based on LS mean difference using ANCOVA where treatment as fixed effect, baseline as the covariate; Test type: Superiority or Other; p = 0.2288, ANCOVA; LS mean difference = 3.51, 90% CI 2-sided [-1.31 to 8.34], Standard Error of Mean 2.897
Statistical Analysis 12: Comparison: PF-04171327 25 mg + Placebo vs Prednisone 5 mg + Placebo; [analysis description as in outcome 9, analysis 11]; Test type: Superiority or Other; p = 0.0980, ANCOVA; LS mean difference = 4.77, 90% CI 2-sided [0.03 to 9.50], Standard Error of Mean 2.844
Statistical Analysis 13: Comparison: PF-04171327 10 mg + Placebo vs Placebo; [analysis description as in outcome 9, analysis 11]; Test type: Superiority or Other; p = 0.0637, ANCOVA; LS mean difference = 5.54, 90% CI 2-sided [0.64 to 10.43], Standard Error of Mean 2.941
Statistical Analysis 14: Comparison: PF-04171327 25 mg + Placebo vs Placebo; [analysis description as in outcome 9, analysis 11]; Test type: Superiority or Other; p = 0.0190, ANCOVA; LS mean difference = 6.79, 90% CI 2-sided [2.07 to 11.50], Standard Error of Mean 2.831
Statistical Analysis 15: Comparison: Prednisone 5 mg + Placebo vs Placebo; [analysis description as in outcome 9, analysis 11]; Test type: Superiority or Other; p = 0.4886, ANCOVA; LS mean difference = 2.02, 90% CI 2-sided [-2.81 to 6.86], Standard Error of Mean 2.903
Statistical Analysis 16: Comparison: PF-04171327 10 mg + Placebo vs Prednisone 5 mg + Placebo; General health at D14: Treatment difference and its corresponding 90% CI was based on LS mean difference using ANCOVA where treatment as fixed effect, baseline as the covariate; Test type: Superiority or Other; p = 0.9951, ANCOVA; LS mean difference = 0.01, 90% CI 2-sided [-3.12 to 3.14], Standard Error of Mean 1.879
Statistical Analysis 17: Comparison: PF-04171327 25 mg + Placebo vs Prednisone 5 mg + Placebo; [analysis description as in outcome 9, analysis 16]; Test type: Superiority or Other; p = 0.4721, ANCOVA; LS mean difference = 1.31, 90% CI 2-sided [-1.71 to 4.34], Standard Error of Mean 1.818
Statistical Analysis 18: Comparison: PF-04171327 10 mg + Placebo vs Placebo; [analysis description as in outcome 9, analysis 16]; Test type: Superiority or Other; p = 0.6835, ANCOVA; LS mean difference = -0.77, 90% CI 2-sided [-3.90 to 2.36], Standard Error of Mean 1.879
Statistical Analysis 19: Comparison: PF-04171327 25 mg + Placebo vs Placebo; [analysis description as in outcome 9, analysis 16]; Test type: Superiority or Other; p = 0.7701, ANCOVA; LS mean difference = 0.53, 90% CI 2-sided [-2.49 to 3.56], Standard Error of Mean 1.818
Statistical Analysis 20: Comparison: Prednisone 5 mg + Placebo vs Placebo; [analysis description as in outcome 9, analysis 16]; Test type: Superiority or Other; p = 0.6710, ANCOVA; LS mean difference = -0.78, 90% CI 2-sided [-3.83 to 2.27], Standard Error of Mean 1.831
Statistical Analysis 21: Comparison: PF-04171327 10 mg + Placebo vs Prednisone 5 mg + Placebo; Vitality at D14: Treatment difference and its corresponding 90% CI was based on LS mean difference using ANCOVA where treatment as fixed effect, baseline as the covariate; Test type: Superiority or Other; p = 0.2886, ANCOVA; LS mean difference = 3.02, 90% CI 2-sided [-1.69 to 7.73], Standard Error of Mean 2.827
Statistical Analysis 22: Comparison: PF-04171327 25 mg + Placebo vs Prednisone 5 mg + Placebo; [analysis description as in outcome 9, analysis 21]; Test type: Superiority or Other; p = 0.1340, ANCOVA; LS mean difference = 4.22, 90% CI 2-sided [-0.42 to 8.86], Standard Error of Mean 2.784
Statistical Analysis 23: Comparison: PF-04171327 10 mg + Placebo vs Placebo; [analysis description as in outcome 9, analysis 21]; Test type: Superiority or Other; p = 0.2563, ANCOVA; LS mean difference = 3.24, 90% CI 2-sided [-1.48 to 7.95], Standard Error of Mean 2.830
Statistical Analysis 24: Comparison: PF-04171327 25 mg + Placebo vs Placebo; [analysis description as in outcome 9, analysis 21]; Test type: Superiority or Other; p = 0.1138, ANCOVA; LS mean difference = 4.43, 90% CI 2-sided [-0.18 to 9.05], Standard Error of Mean 2.771
Statistical Analysis 25: Comparison: Prednisone 5 mg + Placebo vs Placebo; [analysis description as in outcome 9, analysis 21]; Test type: Superiority or Other; p = 0.9386, ANCOVA; LS mean difference = 0.22, 90% CI 2-sided [-4.44 to 4.87], Standard Error of Mean 2.793
Statistical Analysis 26: Comparison: PF-04171327 10 mg + Placebo vs Prednisone 5 mg + Placebo; Social functioning at D14: Treatment difference and its corresponding 90% CI was based on LS mean difference using ANCOVA where treatment as fixed effect, baseline as the covariate; Test type: Superiority or Other; p = 0.8814, ANCOVA; LS mean difference = 0.40, 90% CI 2-sided [-4.09 to 4.90], Standard Error of Mean 2.701
Statistical Analysis 27: Comparison: PF-04171327 25 mg + Placebo vs Prednisone 5 mg + Placebo; [analysis description as in outcome 9, analysis 26]; Test type: Superiority or Other; p = 0.1363, ANCOVA; LS mean difference = 3.98, 90% CI 2-sided [-0.42 to 8.37], Standard Error of Mean 2.640
Statistical Analysis 28: Comparison: PF-04171327 10 mg + Placebo vs Placebo; [analysis description as in outcome 9, analysis 26]; Test type: Superiority or Other; p = 0.7864, ANCOVA; LS mean difference = 0.73, 90% CI 2-sided [-3.74 to 5.20], Standard Error of Mean 2.682
Statistical Analysis 29: Comparison: PF-04171327 25 mg + Placebo vs Placebo; [analysis description as in outcome 9, analysis 26]; Test type: Superiority or Other; p = 0.1048, ANCOVA; LS mean difference = 4.30, 90% CI 2-sided [-0.06 to 8.66], Standard Error of Mean 2.619
Statistical Analysis 30: Comparison: Prednisone 5 mg + Placebo vs Placebo; [analysis description as in outcome 9, analysis 26]; Test type: Superiority or Other; p = 0.9024, ANCOVA; LS mean difference = 0.33, 90% CI 2-sided [-4.08 to 4.73], Standard Error of Mean 2.643
Statistical Analysis 31: Comparison: PF-04171327 10 mg + Placebo vs Prednisone 5 mg + Placebo; Role emotional at D14: Treatment difference and its corresponding 90% CI was based on LS mean difference using ANCOVA where treatment as fixed effect, baseline as the covariate; Test type: Superiority or Other; p = 0.4954, ANCOVA; LS mean difference = 2.62, 90% CI 2-sided [-3.74 to 8.98], Standard Error of Mean 3.819
Statistical Analysis 32: Comparison: PF-04171327 25 mg + Placebo vs Prednisone 5 mg + Placebo; [analysis description as in outcome 9, analysis 31]; Test type: Superiority or Other; p = 0.1729, ANCOVA; LS mean difference = 5.14, 90% CI 2-sided [-1.08 to 11.36], Standard Error of Mean 3.735
Statistical Analysis 33: Comparison: PF-04171327 10 mg + Placebo vs Placebo; [analysis description as in outcome 9, analysis 31]; Test type: Superiority or Other; p = 0.5650, ANCOVA; LS mean difference = 2.21, 90% CI 2-sided [-4.15 to 8.57], Standard Error of Mean 3.820
Statistical Analysis 34: Comparison: PF-04171327 25 mg + Placebo vs Placebo; [analysis description as in outcome 9, analysis 31]; Test type: Superiority or Other; p = 0.2087, ANCOVA; LS mean difference = 4.73, 90% CI 2-sided [-1.48 to 10.94], Standard Error of Mean 3.730
Statistical Analysis 35: Comparison: Prednisone 5 mg + Placebo vs Placebo; [analysis description as in outcome 9, analysis 31]; Test type: Superiority or Other; p = 0.9139, ANCOVA; LS mean difference = -0.41, 90% CI 2-sided [-6.69 to 5.87], Standard Error of Mean 3.771
Statistical Analysis 36: Comparison: PF-04171327 10 mg + Placebo vs Prednisone 5 mg + Placebo; Mental health at D14: Treatment difference and its corresponding 90% CI was based on LS mean difference using ANCOVA where treatment as fixed effect, baseline as the covariate; Test type: Superiority or Other; p = 0.6559, ANCOVA; LS mean difference = 1.51, 90% CI 2-sided [-4.11 to 7.12], Standard Error of Mean 3.371
Statistical Analysis 37: Comparison: PF-04171327 25 mg + Placebo vs Prednisone 5 mg + Placebo; [analysis description as in outcome 9, analysis 36]; Test type: Superiority or Other; p = 0.7304, ANCOVA; LS mean difference = 1.15, 90% CI 2-sided [-4.37 to 6.67], Standard Error of Mean 3.315
Statistical Analysis 38: Comparison: PF-04171327 10 mg + Placebo vs Placebo; [analysis description as in outcome 9, analysis 36]; Test type: Superiority or Other; p = 0.1729, ANCOVA; LS mean difference = 4.64, 90% CI 2-sided [-0.98 to 10.25], Standard Error of Mean 3.369
Statistical Analysis 39: Comparison: PF-04171327 25 mg + Placebo vs Placebo; [analysis description as in outcome 9, analysis 36]; Test type: Superiority or Other; p = 0.2038, ANCOVA; LS mean difference = 4.27, 90% CI 2-sided [-1.28 to 9.83], Standard Error of Mean 3.335
Statistical Analysis 40: Comparison: Prednisone 5 mg + Placebo vs Placebo; [analysis description as in outcome 9, analysis 36]; Test type: Superiority or Other; p = 0.3503, ANCOVA; LS mean difference = 3.13, 90% CI 2-sided [-2.41 to 8.67], Standard Error of Mean 3.328
Statistical Analysis 41: Comparison: PF-04171327 10 mg + Placebo vs Prednisone 5 mg + Placebo; Physical component at D14: Treatment difference and its corresponding 90% CI was based on LS mean difference using ANCOVA where treatment as fixed effect, baseline as the covariate; Test type: Superiority or Other; p = 0.8875, ANCOVA; LS mean difference = 0.29, 90% CI 2-sided [-3.06 to 3.63], Standard Error of Mean 2.010
Statistical Analysis 42: Comparison: PF-04171327 25 mg + Placebo vs Prednisone 5 mg + Placebo; [analysis description as in outcome 9, analysis 41]; Test type: Superiority or Other; p = 0.3203, ANCOVA; LS mean difference = 1.97, 90% CI 2-sided [-1.31 to 5.25], Standard Error of Mean 1.971
Statistical Analysis 43: Comparison: PF-04171327 10 mg + Placebo vs Placebo; [analysis description as in outcome 9, analysis 41]; Test type: Superiority or Other; p = 0.5232, ANCOVA; LS mean difference = 1.31, 90% CI 2-sided [-2.09 to 4.72], Standard Error of Mean 2.046
Statistical Analysis 44: Comparison: PF-04171327 25 mg + Placebo vs Placebo; [analysis description as in outcome 9, analysis 41]; Test type: Superiority or Other; p = 0.1324, ANCOVA; LS mean difference = 3.00, 90% CI 2-sided [-0.28 to 6.28], Standard Error of Mean 1.971
Statistical Analysis 45: Comparison: Prednisone 5 mg + Placebo vs Placebo; [analysis description as in outcome 9, analysis 41]; Test type: Superiority or Other; p = 0.6134, ANCOVA; LS mean difference = 1.03, 90% CI 2-sided [-2.34 to 4.40], Standard Error of Mean 2.024
Statistical Analysis 46: Comparison: PF-04171327 10 mg + Placebo vs Prednisone 5 mg + Placebo; Mental component at D14: Treatment difference and its corresponding 90% CI was based on LS mean difference using ANCOVA where treatment as fixed effect, baseline as the covariate; Test type: Superiority or Other; p = 0.5059, ANCOVA; LS mean difference = 2.26, 90% CI 2-sided [-3.38 to 7.91], Standard Error of Mean 3.387
Statistical Analysis 47: Comparison: PF-04171327 25 mg + Placebo vs Prednisone 5 mg + Placebo; [analysis description as in outcome 9, analysis 46]; Test type: Superiority or Other; p = 0.3042, ANCOVA; LS mean difference = 3.44, 90% CI 2-sided [-2.10 to 8.99], Standard Error of Mean 3.329
Statistical Analysis 48: Comparison: PF-04171327 10 mg + Placebo vs Placebo; [analysis description as in outcome 9, analysis 46]; Test type: Superiority or Other; p = 0.3519, ANCOVA; LS mean difference = 3.18, 90% CI 2-sided [-2.47 to 8.82], Standard Error of Mean 3.390
Statistical Analysis 49: Comparison: PF-04171327 25 mg + Placebo vs Placebo; [analysis description as in outcome 9, analysis 46]; Test type: Superiority or Other; p = 0.1966, ANCOVA; LS mean difference = 4.36, 90% CI 2-sided [-1.21 to 9.92], Standard Error of Mean 3.342
Statistical Analysis 50: Comparison: Prednisone 5 mg + Placebo vs Placebo; [analysis description as in outcome 9, analysis 46]; Test type: Superiority or Other; p = 0.7860, ANCOVA; LS mean difference = 0.91, 90% CI 2-sided [-4.66 to 6.48], Standard Error of Mean 3.345

10. Secondary Outcome: Change From Baseline in Disease Activity Score Based on 28-Joints Count and C-Reactive Protein (3 Variables) (DAS28-3 [CRP]) at Day 7, 14 and 42
Description: DAS28-3 (CRP) was calculated from the swollen joint count and tender joint count using the 28 joints count and CRP (normal range of CRP is <10 mg/L, decrease in the level of CRP indicates reduction in inflammation). Total DAS28-3 (CRP) score range: 0 (least severe) to 9.4 (most severe), higher scores indicate more disease activity.
Time Frame: Baseline, Day 7, 14, 42
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-04171327 10 mg + Placebo | PF-04171327 25 mg + Placebo | Prednisone 5 mg + Placebo | Placebo
Number analyzed (Participants) | 21 | 22 | 21 | 22
units on a scale
  Baseline | 5.80 (0.731) | 5.87 (0.674) | 5.59 (0.666) | 5.72 (0.706)
  Change at Day 7: number analyzed (Participants) | 20 | 21 | 21 | 21
  Change at Day 7 | -1.07 (0.800) | -1.51 (0.845) | -0.55 (0.632) | -0.50 (0.609)
  Change at Day 14: number analyzed (Participants) | 18 | 21 | 20 | 21
  Change at Day 14 | -1.57 (0.749) | -2.01 (1.178) | -0.92 (0.994) | -0.87 (0.798)
  Change at Day 42: number analyzed (Participants) | 19 | 21 | 20 | 21
  Change at Day 42 | -0.81 (1.007) | -1.26 (1.199) | -1.17 (0.949) | -1.12 (1.005)
Statistical Analysis 1: Comparison: PF-04171327 10 mg + Placebo vs Prednisone 5 mg + Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.1090, MMRM; LS mean difference = -0.46, 90% CI 2-sided [-0.93 to 0.01], Standard Error of Mean 0.286
Statistical Analysis 2: Comparison: PF-04171327 25 mg + Placebo vs Prednisone 5 mg + Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0014, MMRM; LS mean difference = -0.91, 90% CI 2-sided [-1.38 to -0.45], Standard Error of Mean 0.282
Statistical Analysis 3: Comparison: PF-04171327 10 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0506, MMRM; LS mean difference = -0.56, 90% CI 2-sided [-1.03 to -0.09], Standard Error of Mean 0.284
Statistical Analysis 4: Comparison: PF-04171327 25 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0004, MMRM; LS mean difference = -1.01, 90% CI 2-sided [-1.48 to -0.55], Standard Error of Mean 0.280
Statistical Analysis 5: Comparison: Prednisone 5 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.7272, MMRM; LS mean difference = -0.10, 90% CI 2-sided [-0.56 to 0.37], Standard Error of Mean 0.281
Statistical Analysis 6: Comparison: PF-04171327 10 mg + Placebo vs Prednisone 5 mg + Placebo; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.0604, MMRM; LS mean difference = -0.56, 90% CI 2-sided [-1.05 to -0.07], Standard Error of Mean 0.296
Statistical Analysis 7: Comparison: PF-04171327 25 mg + Placebo vs Prednisone 5 mg + Placebo; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.0003, MMRM; LS mean difference = -1.06, 90% CI 2-sided [-1.53 to -0.59], Standard Error of Mean 0.285
Statistical Analysis 8: Comparison: PF-04171327 10 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.0377, MMRM; LS mean difference = -0.61, 90% CI 2-sided [-1.09 to -0.13], Standard Error of Mean 0.291
Statistical Analysis 9: Comparison: PF-04171327 25 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.0001, MMRM; LS mean difference = -1.11, 90% CI 2-sided [-1.57 to -0.65], Standard Error of Mean 0.280
Statistical Analysis 10: Comparison: Prednisone 5 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.8612, MMRM; LS mean difference = -0.05, 90% CI 2-sided [-0.52 to 0.42], Standard Error of Mean 0.284
Statistical Analysis 11: Comparison: PF-04171327 10 mg + Placebo vs Prednisone 5 mg + Placebo; [analysis description as in outcome 2, analysis 11]; Test type: Superiority or Other; p = 0.1330, MMRM; LS mean difference = 0.44, 90% CI 2-sided [-0.04 to 0.93], Standard Error of Mean 0.292
Statistical Analysis 12: Comparison: PF-04171327 25 mg + Placebo vs Prednisone 5 mg + Placebo; [analysis description as in outcome 2, analysis 11]; Test type: Superiority or Other; p = 0.8542, MMRM; LS mean difference = -0.05, 90% CI 2-sided [-0.52 to 0.42], Standard Error of Mean 0.285
Statistical Analysis 13: Comparison: PF-04171327 10 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 11]; Test type: Superiority or Other; p = 0.2339, MMRM; LS mean difference = 0.34, 90% CI 2-sided [-0.13 to 0.82], Standard Error of Mean 0.288
Statistical Analysis 14: Comparison: PF-04171327 25 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 11]; Test type: Superiority or Other; p = 0.5927, MMRM; LS mean difference = -0.15, 90% CI 2-sided [-0.61 to 0.31], Standard Error of Mean 0.280
Statistical Analysis 15: Comparison: Prednisone 5 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 11]; Test type: Superiority or Other; p = 0.7304, MMRM; LS mean difference = -0.10, 90% CI 2-sided [-0.57 to 0.37], Standard Error of Mean 0.284

11. Secondary Outcome: Change From Baseline in Disease Activity Score Based on 28-Joints Count and C-Reactive Protein (4 Variables) (DAS28-4 [CRP]) at Day 7
Description: DAS28-4 (CRP) examines progression or improvement of RA. It was assessed from SJC and TJC using the 28 joints count, CRP (normal range of CRP is <10 mg/L, decrease in the level of CRP indicates reduction in inflammation) and PGA of disease activity (participant global assessment of diseases condition scores ranging from 0 [very well condition] to 100 [very poor condition], higher scores indicated greater affectation due to disease activity). Total DAS28-4 (CRP) transformed score range: 0 (least severe) to 10 (most severe), higher scores indicate more severe disease activity. DAS28-4 (CRP) scores: <=3.2 implied low disease activity; >3.2 to 5.1 implied moderate to high disease activity.
Time Frame: Baseline, Day 7
Population: FAS included all randomized participants who received at least 1 dose of the randomized investigational drug. Here, 'Number of Participants analyzed' signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-04171327 10 mg + Placebo | PF-04171327 25 mg + Placebo | Prednisone 5 mg + Placebo | Placebo
Number analyzed (Participants) | 20 | 21 | 21 | 21
units on a scale | -1.21 (0.889) | -1.63 (1.034) | -0.67 (0.639) | -0.55 (0.697)
Statistical Analysis 1: Comparison: PF-04171327 10 mg + Placebo vs Prednisone 5 mg + Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0956, MMRM; LS mean difference = -0.49, 90% CI 2-sided [-0.97 to -0.01], Standard Error of Mean 0.290
Statistical Analysis 2: Comparison: PF-04171327 25 mg + Placebo vs Prednisone 5 mg + Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0016, MMRM; LS mean difference = -0.93, 90% CI 2-sided [-1.40 to -0.45], Standard Error of Mean 0.286
Statistical Analysis 3: Comparison: PF-04171327 10 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0258, MMRM; LS mean difference = -0.65, 90% CI 2-sided [-1.13 to -0.17], Standard Error of Mean 0.287
Statistical Analysis 4: Comparison: PF-04171327 25 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0002, MMRM; LS mean difference = -1.09, 90% CI 2-sided [-1.56 to -0.62], Standard Error of Mean 0.283
Statistical Analysis 5: Comparison: Prednisone 5 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.5692, MMRM; LS mean difference = -0.16, 90% CI [-0.63 to 0.31], Standard Error of Mean 0.284

12. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 20% (ACR20) Response at Day 7 and 14
Description: ACR20 responder: participants who achieved at =20% improvement in tender and swollen 28-joints count, and >=20% improvement in at least 3 of the following 5 measures: 1) participant's assessment of arthritis pain (participant's self-assessed severity of arthritis pain, score range from 0[no pain] to 100[most severe pain], higher scores=more pain), 2) PGA of arthritis (participant's assessed overall arthritis activity, score range from 0[no arthritis] to 100[extreme arthritis], higher scores=higher degree of arthritis), 3) PhGA of arthritis (physician rated severity of participants overall arthritis activity, score range from 0[no arthritis] to 100[extreme arthritis], higher scores=higher degree of arthritis), 4) HAQ-DI (assessment of functional disability, score range from 0[no difficulty] to 3[extreme difficulty], higher scores=more functional limitation) and 5) CRP (assessment of inflammation, normal range of CRP is <10 mg/L, decrease in the level of CRP=reduction in inflammation).
Time Frame: Day 7, 14
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PF-04171327 10 mg + Placebo | PF-04171327 25 mg + Placebo | Prednisone 5 mg + Placebo | Placebo
Number analyzed (Participants) | 21 | 22 | 21 | 22
percentage of participants
  Day 7: number analyzed (Participants) | 21 | 21 | 21 | 21
  Day 7 | 28.57 | 52.38 | 14.29 | 27.27
  Day 14: number analyzed (Participants) | 18 | 21 | 20 | 21
  Day 14 | 55.56 | 66.67 | 45.00 | 38.10
Statistical Analysis 1: Comparison: PF-04171327 10 mg + Placebo vs Prednisone 5 mg + Placebo; Day 7; Test type: Superiority or Other; p = 0.1460, Barnard exact test; Difference in percentage = 14.29, 90% CI 2-sided [-8.65 to 35.98]
Statistical Analysis 2: Comparison: PF-04171327 25 mg + Placebo vs Prednisone 5 mg + Placebo; Day 7; Test type: Superiority or Other; p = 0.0052, Barnard exact test; Difference in percentage = 38.10, 90% CI 2-sided [12.25 to 59.46]
Statistical Analysis 3: Comparison: PF-04171327 10 mg + Placebo vs Placebo; Day 7; Test type: Superiority or Other; p = 0.5094, Barnard exact test; Difference in percentage = 1.30, 90% CI 2-sided [-22.00 to 24.66]
Statistical Analysis 4: Comparison: PF-04171327 25 mg + Placebo vs Placebo; Day 7; Test type: Superiority or Other; p = 0.0551, Barnard exact test; Difference in percentage = 25.11, 90% CI 2-sided [-0.69 to 48.34]
Statistical Analysis 5: Comparison: Prednisone 5 mg + Placebo vs Placebo; Day 7; Test type: Superiority or Other; p = 0.9999, Barnard exact test; Difference in percentage = -12.99, 90% CI 2-sided [-34.09 to 8.78]
Statistical Analysis 6: Comparison: PF-04171327 10 mg + Placebo vs Prednisone 5 mg + Placebo; Day 14; Test type: Superiority or Other; p = 0.3027, Barnard-Exact test; Difference in percentage = 10.56, 90% CI 2-sided [-17.18 to 37.67]
Statistical Analysis 7: Comparison: PF-04171327 25 mg + Placebo vs Prednisone 5 mg + Placebo; Day 14; Test type: Superiority or Other; p = 0.1074, Barnard-Exact test; Difference in percentage = 21.67, 90% CI 2-sided [-6.24 to 46.16]
Statistical Analysis 8: Comparison: PF-04171327 10 mg + Placebo vs Placebo; Day 14; Test type: Superiority or Other; p = 0.2340, Barnard-Exact test; Difference in percentage = 17.46, 90% CI 2-sided [-10.08 to 43.70]
Statistical Analysis 9: Comparison: PF-04171327 25 mg + Placebo vs Placebo; Day 14; Test type: Superiority or Other; p = 0.0442, Barnard-Exact test; Difference in percentage = 28.57, 90% CI 2-sided [0.91 to 53.07]
Statistical Analysis 10: Comparison: Prednisone 5 mg + Placebo vs Placebo; Day 14; Test type: Superiority or Other; p = 0.3813, Barnard-Exact test; Difference in percentage = 6.90, 90% CI 2-sided [-19.82 to 32.92]

13. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 50% (ACR50) Response at Day 7 and 14
Description: ACR50 responder: participants who achieved at =50% improvement in tender and swollen 28-joints count, and >=50% improvement in at least 3 of the following 5 measures: 1) participant's assessment of arthritis pain (participant's self-assessed severity of arthritis pain, score range from 0[no pain] to 100[most severe pain], higher scores=more pain), 2) PGA of arthritis (participant's assessed overall arthritis activity, score range from 0[no arthritis] to 100[extreme arthritis], higher scores=higher degree of arthritis), 3) PhGA of arthritis (physician rated severity of participants overall arthritis activity, score range from 0[no arthritis] to 100[extreme arthritis], higher scores=higher degree of arthritis), 4) HAQ-DI (assessment of functional disability, score range from 0[no difficulty] to 3[extreme difficulty], higher scores=more functional limitation) and 5) CRP (assessment of inflammation, normal range of CRP is <10 mg/L, decrease in the level of CRP=reduction in inflammation).
Time Frame: Day 7, 14
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PF-04171327 10 mg + Placebo | PF-04171327 25 mg + Placebo | Prednisone 5 mg + Placebo | Placebo
Number analyzed (Participants) | 21 | 22 | 21 | 22
percentage of participants
  Day 7: number analyzed (Participants) | 21 | 21 | 21 | 22
  Day 7 | 9.52 | 19.05 | 0.00 | 0.00
  Day 14: number analyzed (Participants) | 18 | 21 | 20 | 21
  Day 14 | 22.22 | 47.62 | 20.00 | 14.29
Statistical Analysis 1: Comparison: PF-04171327 10 mg + Placebo vs Prednisone 5 mg + Placebo; Day 7; Test type: Superiority or Other; p = 0.1017, Barnard exact test; Difference in percentage = 9.52, 90% CI 2-sided [-3.90 to 27.09]
Statistical Analysis 2: Comparison: PF-04171327 25 mg + Placebo vs Prednisone 5 mg + Placebo; Day 7; Test type: Superiority or Other; p = 0.0218, Barnard exact test; Difference in percentage = 19.05, 90% CI 2-sided [4.49 to 38.44]
Statistical Analysis 3: Comparison: PF-04171327 10 mg + Placebo vs Placebo; Day 7; Test type: Superiority or Other; p = 0.1082, Barnard exact test; Difference in percentage = 9.52, 90% CI 2-sided [-3.71 to 27.06]
Statistical Analysis 4: Comparison: PF-04171327 25 mg + Placebo vs Placebo; Day 7; Test type: Superiority or Other; p = 0.0166, Barnard exact test; Difference in percentage = 19.05, 90% CI 2-sided [4.81 to 38.44]
Statistical Analysis 5: Comparison: PF-04171327 10 mg + Placebo vs Prednisone 5 mg + Placebo; Day 14; Test type: Superiority or Other; p = 0.4776, Barnard exact test; Difference in percentage = 2.22, 90% CI 2-sided [-21.61 to 25.87]
Statistical Analysis 6: Comparison: PF-04171327 25 mg + Placebo vs Prednisone 5 mg + Placebo; Day 14; Test type: Superiority or Other; p = 0.0347, Barnard exact test; Difference in percentage = 27.62, 90% CI 2-sided [2.53 to 50.78]
Statistical Analysis 7: Comparison: PF-04171327 10 mg + Placebo vs Placebo; Day 14; Test type: Superiority or Other; p = 0.3343, Barnard exact test; Difference in percentage = 7.94, 90% CI 2-sided [-13.71 to 31.59]
Statistical Analysis 8: Comparison: PF-04171327 25 mg + Placebo vs Placebo; Day 14; Test type: Superiority or Other; p = 0.0117, Barnard exact test; Difference in percentage = 33.33, 90% CI 2-sided [8.35 to 55.00]
Statistical Analysis 9: Comparison: Prednisone 5 mg + Placebo vs Placebo; Day 14; Test type: Superiority or Other; p = 0.3720, Barnard exact test; Difference in percentage = 5.71, 90% CI 2-sided [-15.86 to 27.04]

14. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 70% (ACR70) Response at Day 7 and 14
Description: ACR70 responder: participants who achieved at =70% improvement in tender and swollen 28-joints count, and >=70% improvement in at least 3 of the following 5 measures: 1) participant's assessment of arthritis pain (participant's self-assessed severity of arthritis pain, score range from 0[no pain] to 100[most severe pain], higher scores=more pain), 2) PGA of arthritis (participant's assessed overall arthritis activity, score range from 0[no arthritis] to 100[extreme arthritis], higher scores=higher degree of arthritis), 3) PhGA of arthritis (physician rated severity of participants overall arthritis activity, score range from 0[no arthritis] to 100[extreme arthritis], higher scores=higher degree of arthritis), 4) HAQ-DI (assessment of functional disability, score range from 0[no difficulty] to 3[extreme difficulty], higher scores=more functional limitation) and 5) CRP (assessment of inflammation, normal range of CRP is <10 mg/L, decrease in the level of CRP=reduction in inflammation).
Time Frame: Day 7, 14
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | PF-04171327 10 mg + Placebo | PF-04171327 25 mg + Placebo | Prednisone 5 mg + Placebo | Placebo
Number analyzed (Participants) | 21 | 22 | 21 | 22
percentage of participants
  Day 7: number analyzed (Participants) | 21 | 21 | 21 | 22
  Day 7 | 4.76 | 4.76 | 0.00 | 0.00
  Day 14: number analyzed (Participants) | 18 | 21 | 20 | 21
  Day 14 | 0.00 | 14.29 | 0.00 | 0.00
Statistical Analysis 1: Comparison: PF-04171327 10 mg + Placebo vs Prednisone 5 mg + Placebo; Day 7; Test type: Superiority or Other; p = 0.2630, Barnard exact test; Difference in percentage = 4.76, 90% CI 2-sided [-8.61 to 20.67]
Statistical Analysis 2: Comparison: PF-04171327 25 mg + Placebo vs Prednisone 5 mg + Placebo; Day 7; Test type: Superiority or Other; p = 0.2630, Barnard exact test; Difference in percentage = 4.76, 90% CI 2-sided [-8.61 to 20.67]
Statistical Analysis 3: Comparison: PF-04171327 10 mg + Placebo vs Placebo; Day 7; Test type: Superiority or Other; p = 0.2539, Barnard exact test; Difference in percentage = 4.76, 90% CI 2-sided [-7.51 to 20.67]
Statistical Analysis 4: Comparison: PF-04171327 25 mg + Placebo vs Placebo; Day 7; Test type: Superiority or Other; p = 0.2539, Barnard exact test; Difference in percentage = 4.76, 90% CI 2-sided [-7.51 to 20.67]
Statistical Analysis 5: Comparison: PF-04171327 25 mg + Placebo vs Prednisone 5 mg + Placebo; Day 14; Test type: Superiority or Other; p = 0.0477, Barnard exact test; Difference in percentage = 14.29, 90% CI 2-sided [0.23 to 32.92]
Statistical Analysis 6: Comparison: PF-04171327 25 mg + Placebo vs Placebo; Day 14; Test type: Superiority or Other; p = 0.0442, Barnard exact test; Difference in percentage = 14.29, 90% CI 2-sided [0.65 to 32.92]

15. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 31 days after last dose (Day 45) that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Baseline up to Day 45
Population: Safety analysis set included all randomized participants who received at least 1 dose of the randomized investigational drug.
Measure: Number; unit: participants
Arm/Group | PF-04171327 10 mg + Placebo | PF-04171327 25 mg + Placebo | Prednisone 5 mg + Placebo | Placebo
Number analyzed (Participants) | 21 | 22 | 21 | 22
participants
  AE | 8 | 3 | 4 | 12
  SAE | 0 | 0 | 0 | 0

16. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Laboratory Abnormalities
Description: Criteria for laboratory abnormalities: Hematology (hemoglobin, hematocrit <0.8*baseline; platelet count <75 or >700*10^3 per mm^3; leucocytes <2.5 or >17.5*10^3 per mm^3); chemistry (total bilirubin >1.5*upper limit of reference range [ULN]; aspartate aminotransferase, alanine aminotransferase, gamma-glutamyl transpeptidase, alkaline phosphatase, >3.0*ULN; total protein, albumin <0.8*lower limit of reference range [LLN] or >1.2*ULN; blood urea nitrogen [BUN]/urea, creatinine >1.3*ULN; glucose [fasting] <0.6*LLN or >1.5*ULN; uric acid >1.2*ULN; sodium <0.95*LLN or >1.05*ULN; potassium, calcium <0.9*LLN or >1.1*ULN; albumin, total protein <0.8*LLN or >1.2*ULN; urinalysis (urine white blood cell (WBC) =>6/ high power field (hpf); urine red blood cell (RBC) =>6/hpf). Number of participants with clinically significant change from baseline in laboratory abnormalities identified by investigator were reported.
Time Frame: Baseline up to Day 45
Population: as for outcome 15
Measure: Number; unit: participants
Arm/Group | PF-04171327 10 mg + Placebo | PF-04171327 25 mg + Placebo | Prednisone 5 mg + Placebo | Placebo
Number analyzed (Participants) | 21 | 22 | 21 | 22
participants | 0 | 0 | 0 | 0

17. Secondary Outcome: Change From Baseline in Body Weight at Day 7 and 14
Time Frame: Baseline, Day 7, 14
Population: Safety analysis set included all randomized participants who received at least 1 dose of the randomized investigational drug. Here, 'n' signifies those participants who were evaluable at specified time points, respectively.
Measure: Mean (Standard Deviation); unit: kilogram
Arm/Group | PF-04171327 10 mg + Placebo | PF-04171327 25 mg + Placebo | Prednisone 5 mg + Placebo | Placebo
Number analyzed (Participants) | 21 | 22 | 21 | 22
kilogram
  Baseline | 83.7 (17.0) | 74.1 (16.1) | 78.4 (15.4) | 75.0 (17.2)
  Change at Day 7: number analyzed (Participants) | 21 | 21 | 21 | 22
  Change at Day 7 | 0.12 (0.733) | -0.04 (1.256) | -0.02 (1.036) | -0.05 (0.858)
  Change at Day 14: number analyzed (Participants) | 19 | 21 | 20 | 21
  Change at Day 14 | 0.35 (1.064) | 0.20 (1.158) | 0.18 (1.467) | -0.04 (0.903)
Statistical Analysis 1: Comparison: PF-04171327 10 mg + Placebo vs Prednisone 5 mg + Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.5403, MMRM; LS mean difference = 0.20, 90% CI 2-sided [-0.34 to 0.75], Standard Error of Mean 0.330
Statistical Analysis 2: Comparison: PF-04171327 25 mg + Placebo vs Prednisone 5 mg + Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.8374, MMRM; LS mean difference = -0.07, 90% CI 2-sided [-0.61 to 0.48], Standard Error of Mean 0.330
Statistical Analysis 3: Comparison: PF-04171327 10 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.4305, MMRM; LS mean difference = 0.26, 90% CI 2-sided [-0.28 to 0.80], Standard Error of Mean 0.329
Statistical Analysis 4: Comparison: PF-04171327 25 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.9733, MMRM; LS mean difference = -0.01, 90% CI 2-sided [-0.55 to 0.53], Standard Error of Mean 0.325
Statistical Analysis 5: Comparison: Prednisone 5 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.8613, MMRM; LS mean difference = 0.06, 90% CI 2-sided [-0.48 to 0.60], Standard Error of Mean 0.325
Statistical Analysis 6: Comparison: PF-04171327 10 mg + Placebo vs Prednisone 5 mg + Placebo; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.5245, MMRM; LS mean difference = 0.22, 90% CI 2-sided [-0.35 to 0.78], Standard Error of Mean 0.341
Statistical Analysis 7: Comparison: PF-04171327 25 mg + Placebo vs Prednisone 5 mg + Placebo; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.8917, MMRM; LS mean difference = -0.05, 90% CI 2-sided [-0.60 to 0.51], Standard Error of Mean 0.334
Statistical Analysis 8: Comparison: PF-04171327 10 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.1695, MMRM; LS mean difference = 0.47, 90% CI 2-sided [-0.09 to 1.03], Standard Error of Mean 0.339
Statistical Analysis 9: Comparison: PF-04171327 25 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.5339, MMRM; LS mean difference = 0.20, 90% CI 2-sided [-0.34 to 0.75], Standard Error of Mean 0.329
Statistical Analysis 10: Comparison: Prednisone 5 mg + Placebo vs Placebo; [analysis description as in outcome 2, analysis 6]; Test type: Superiority or Other; p = 0.4520, MMRM; LS mean difference = 0.25, 90% CI 2-sided [-0.30 to 0.80], Standard Error of Mean 0.332

18. Secondary Outcome: Number of Participants With Clinically Significant Vital Signs Abnormalities
Description: Following parameters were analyzed for examination of vital signs: systolic and diastolic blood pressure, heart rate and body temperature. Vital sign measurements were performed with the participant in the seated position. Clinical significance vital sign abnormality was determined by investigator.
Time Frame: Baseline up to Day 45
Population: as for outcome 15
Measure: Number; unit: participants
Arm/Group | PF-04171327 10 mg + Placebo | PF-04171327 25 mg + Placebo | Prednisone 5 mg + Placebo | Placebo
Number analyzed (Participants) | 21 | 22 | 21 | 22
participants | 0 (6.55) | 0 (7.78) | 0 (7.30) | 0 (7.54)

19. Secondary Outcome: Number of Participants With Clinically Significant Electrocardiogram (ECG) Abnormalities
Description: Clinically significant ECG findings included PR interval >=300 milliseconds (msec) or >=25% increase from baseline (if baseline PR interval >200 msec) or >=50% increase (if baseline PR interval less than or equal to [<=] 200 msec); QRS interval >=200 msec or >=25% increase from baseline (if baseline PR interval >100 msec) or >=50% increase (if baseline PR interval <= 100 msec); QT interval >=500 msec, corrected QT interval >=500 msec.
Time Frame: Baseline up to Day 45
Population: as for outcome 15
Measure: Number; unit: participants
Arm/Group | PF-04171327 10 mg + Placebo | PF-04171327 25 mg + Placebo | Prednisone 5 mg + Placebo | Placebo
Number analyzed (Participants) | 21 | 22 | 21 | 22
participants | 0 | 0 | 0 | 0

20. Secondary Outcome: Plasma Concentration of PF-00251802 Versus Time Summary on Day 7 and Day 14
Description: Plasma concentration of PF-00251802 versus time summary, a metabolite of PF-04171327 was reported in this outcome measure.
Time Frame: 0, 1, 2, 3 and 4 hours post-dose on Day 7, 14
Population: Analysis set included all randomized participants who received at least 1 dose of PF-04171327. Here, 'Number of Participants analyzed' signifies those participants who were evaluable for this outcome measure. Here, 'n' signifies those participants who were evaluable at specified time points, respectively.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | PF-04171327 10 mg + Placebo | PF-04171327 25 mg + Placebo
Number analyzed (Participants) | 19 | 20
nanogram per milliliter (ng/mL)
  Day 7 (0 hour): number analyzed (Participants) | 18 | 19
  Day 7 (0 hour) | 53.07 (21.480) | 136.8 (82.246)
  Day 7 (1 hour): number analyzed (Participants) | 17 | 18
  Day 7 (1 hour) | 90.28 (50.250) | 257.9 (93.716)
  Day 7 (2 hour): number analyzed (Participants) | 17 | 19
  Day 7 (2 hour) | 118.1 (40.314) | 281.3 (73.866)
  Day 7 (3 hour): number analyzed (Participants) | 17 | 19
  Day 7 (3 hour) | 116.3 (42.988) | 230.7 (82.895)
  Day 7 (4 hour): number analyzed (Participants) | 17 | 19
  Day 7 (4 hour) | 107.5 (27.303) | 220.6 (53.416)
  Day 14 (0 hour): number analyzed (Participants) | 18 | 18
  Day 14 (0 hour) | 53.94 (25.382) | 136.3 (53.159)
  Day 14 (1 hour): number analyzed (Participants) | 17 | 18
  Day 14 (1 hour) | 115.7 (64.846) | 216.4 (102.88)
  Day 14 (2 hour): number analyzed (Participants) | 17 | 18
  Day 14 (2 hour) | 133.9 (50.294) | 284.9 (117.38)
  Day 14 (3 hour): number analyzed (Participants) | 17 | 18
  Day 14 (3 hour) | 123.7 (36.720) | 296.6 (119.76)
  Day 14 (4 hour): number analyzed (Participants) | 17 | 18
  Day 14 (4 hour) | 106.3 (28.542) | 243.3 (90.962)

21. Secondary Outcome: Ratio of Apparent Oral Clearance on Day 1 to Day 14 of Methotrexate
Description: Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood. Methotrexate was used as a background therapy by participants.
Time Frame: Pre-dose (0 hour), 1, 2, 3 and 4 hours post-dose
Population: Analysis set included all randomized participants who received at least 1 dose of the randomized investigational drug. Here, 'Number of Participants analyzed' signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Error); unit: ratio
Arm/Group | PF-04171327 10 mg + Placebo | PF-04171327 25 mg + Placebo | Prednisone 5 mg + Placebo | Placebo
Number analyzed (Participants) | 20 | 22 | 21 | 22
ratio | 1.24 (0.12) | 0.98 (0.05) | 1.14 (0.10) | 0.93 (0.07)

22. Secondary Outcome: Change From Baseline in Lymphocyte Counts at Day 1, 7 and 14
Time Frame: Baseline; 1, 2, 3 and 4 hours post-dose on Day 1; 0, 1, 2, 3 and 4 hours post-dose on Day 7 and 14
Population: Analysis set included all randomized participants who received at least 1 dose of the randomized investigational drug. Here, 'n' signifies those participants who were evaluable at specified time points, respectively.
Measure: Mean (Standard Deviation); unit: 10^3 cells per microliter
Arm/Group | PF-04171327 10 mg + Placebo | PF-04171327 25 mg + Placebo | Prednisone 5 mg + Placebo | Placebo
Number analyzed (Participants) | 21 | 22 | 21 | 22
10^3 cells per microliter
  Baseline: number analyzed (Participants) | 21 | 22 | 20 | 22
  Baseline | 1.85 (0.510) | 1.80 (0.856) | 1.68 (0.560) | 1.79 (0.648)
  Change at Day 1: 1 hour: number analyzed (Participants) | 21 | 20 | 20 | 22
  Change at Day 1: 1 hour | -0.01 (0.200) | 0.02 (0.304) | 0.13 (0.344) | 0.04 (0.218)
  Change at Day 1: 2 hour: number analyzed (Participants) | 21 | 19 | 19 | 22
  Change at Day 1: 2 hour | 0.28 (0.315) | 0.05 (0.320) | 0.09 (0.326) | 0.09 (0.231)
  Change at Day 1: 3 hour: number analyzed (Participants) | 20 | 19 | 20 | 22
  Change at Day 1: 3 hour | 0.21 (0.322) | 0.07 (0.328) | 0.10 (0.297) | 0.04 (0.455)
  Change at Day 1: 4 hour: number analyzed (Participants) | 21 | 20 | 18 | 22
  Change at Day 1: 4 hour | 0.28 (0.408) | 0.05 (0.428) | 0.07 (0.244) | 0.03 (0.450)
  Change at Day 7: 0 hour: number analyzed (Participants) | 20 | 21 | 20 | 21
  Change at Day 7: 0 hour | 0.79 (0.384) | 0.83 (0.342) | 0.26 (0.441) | 0.05 (0.270)
  Change at Day 7: 1 hour: number analyzed (Participants) | 19 | 20 | 18 | 20
  Change at Day 7: 1 hour | 0.64 (0.477) | 0.62 (0.438) | 0.13 (0.589) | -0.03 (0.275)
  Change at Day 7: 2 hour: number analyzed (Participants) | 19 | 21 | 19 | 21
  Change at Day 7: 2 hour | 0.76 (0.416) | 0.76 (0.463) | -0.03 (0.505) | 0.10 (0.287)
  Change at Day 7: 3 hour: number analyzed (Participants) | 19 | 21 | 19 | 21
  Change at Day 7: 3 hour | 0.77 (0.465) | 0.85 (0.563) | -0.25 (0.539) | 0.15 (0.345)
  Change at Day 7: 4 hour: number analyzed (Participants) | 19 | 20 | 19 | 20
  Change at Day 7: 4 hour | 0.72 (0.470) | 0.69 (0.478) | -0.23 (0.431) | 0.19 (0.402)
  Change at Day 14: 0 hour: number analyzed (Participants) | 17 | 20 | 17 | 19
  Change at Day 14: 0 hour | 0.89 (0.308) | 0.82 (0.638) | 0.29 (0.492) | -0.07 (0.322)
  Change at Day 14: 1 hour: number analyzed (Participants) | 17 | 20 | 19 | 17
  Change at Day 14: 1 hour | 0.81 (0.425) | 0.66 (0.589) | 0.22 (0.421) | -0.03 (0.294)
  Change at Day 14: 2 hour: number analyzed (Participants) | 17 | 20 | 19 | 17
  Change at Day 14: 2 hour | 0.74 (0.340) | 0.62 (0.680) | -0.03 (0.467) | 0.04 (0.441)
  Change at Day 14: 3 hour: number analyzed (Participants) | 17 | 20 | 18 | 16
  Change at Day 14: 3 hour | 0.81 (0.494) | 0.75 (0.634) | -0.35 (0.397) | 0.20 (0.238)
  Change at Day 14: 4 hour: number analyzed (Participants) | 17 | 20 | 18 | 20
  Change at Day 14: 4 hour | 0.77 (0.428) | 0.57 (0.445) | -0.45 (0.396) | 0.08 (0.268)

23. Secondary Outcome: Change From Baseline in Neutrophil Counts at Day 1, 7 and 14
Time Frame: Baseline; 1, 2, 3 and 4 hours post-dose on Day 1; 0, 1, 2, 3 and 4 hours post-dose on Day 7 and 14
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: 10^3 cells per microliter
Arm/Group | PF-04171327 10 mg + Placebo | PF-04171327 25 mg + Placebo | Prednisone 5 mg + Placebo | Placebo
Number analyzed (Participants) | 21 | 22 | 21 | 22
10^3 cells per microliter
  Baseline: number analyzed (Participants) | 21 | 22 | 20 | 22
  Baseline | 5.43 (2.050) | 5.53 (3.091) | 5.90 (2.127) | 5.03 (2.029)
  Change at Day 1: 1 hour: number analyzed (Participants) | 21 | 20 | 20 | 22
  Change at Day 1: 1 hour | 0.04 (0.799) | 0.42 (0.581) | 0.45 (0.853) | 0.09 (0.534)
  Change at Day 1: 2 hour: number analyzed (Participants) | 21 | 19 | 19 | 22
  Change at Day 1: 2 hour | 0.01 (0.516) | 0.12 (0.621) | 0.38 (1.109) | -0.07 (0.674)
  Change at Day 1: 3 hour: number analyzed (Participants) | 20 | 19 | 20 | 22
  Change at Day 1: 3 hour | -0.06 (0.638) | 0.49 (1.247) | 0.22 (0.999) | -0.05 (0.812)
  Change at Day 1: 4 hour: number analyzed (Participants) | 21 | 20 | 18 | 22
  Change at Day 1: 4 hour | -0.28 (0.876) | 0.34 (1.625) | -0.03 (0.984) | -0.25 (0.831)
  Change at Day 7: 0 hour: number analyzed (Participants) | 20 | 21 | 20 | 21
  Change at Day 7: 0 hour | 0.16 (1.036) | 0.06 (1.993) | 0.22 (1.401) | -0.21 (1.217)
  Change at Day 7: 1 hour: number analyzed (Participants) | 19 | 20 | 18 | 20
  Change at Day 7: 1 hour | 0.63 (1.145) | 0.21 (1.947) | 0.64 (1.776) | 0.07 (1.202)
  Change at Day 7: 2 hour: number analyzed (Participants) | 19 | 21 | 19 | 21
  Change at Day 7: 2 hour | 0.79 (1.195) | 0.80 (2.278) | 1.66 (1.764) | -0.06 (1.292)
  Change at Day 7: 3 hour: number analyzed (Participants) | 19 | 21 | 19 | 21
  Change at Day 7: 3 hour | 1.19 (1.304) | 1.19 (2.120) | 2.14 (1.828) | -0.13 (1.252)
  Change at Day 7: 4 hour: number analyzed (Participants) | 19 | 20 | 19 | 20
  Change at Day 7: 4 hour | 1.13 (1.320) | 0.84 (2.159) | 2.01 (1.788) | -0.47 (1.352)
  Change at Day 14: 0 hour: number analyzed (Participants) | 17 | 20 | 17 | 19
  Change at Day 14: 0 hour | 0.32 (0.954) | 0.77 (1.881) | -0.79 (1.291) | -0.11 (1.116)
  Change at Day 14: 1 hour: number analyzed (Participants) | 17 | 20 | 19 | 17
  Change at Day 14: 1 hour | 0.40 (1.114) | 1.00 (1.827) | -0.09 (1.566) | -0.16 (0.731)
  Change at Day 14: 2 hour: number analyzed (Participants) | 17 | 20 | 19 | 17
  Change at Day 14: 2 hour | 0.56 (1.172) | 1.11 (2.097) | 0.74 (1.866) | -0.35 (0.901)
  Change at Day 14: 3 hour: number analyzed (Participants) | 17 | 20 | 18 | 16
  Change at Day 14: 3 hour | 1.10 (1.560) | 1.57 (2.076) | 1.14 (1.788) | -0.41 (1.190)
  Change at Day 14: 4 hour: number analyzed (Participants) | 17 | 20 | 18 | 20
  Change at Day 14: 4 hour | 1.09 (1.559) | 1.39 (2.203) | 1.07 (1.595) | -0.65 (1.347)

24. Secondary Outcome: Change From Baseline in Eosinophil Counts at Day 1, 7 and 14
Time Frame: Baseline; 1, 2, 3 and 4 hours post-dose on Day 1; 0, 1, 2, 3 and 4 hours post-dose on Day 7 and 14
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: 10^3 cells per microliter
Arm/Group | PF-04171327 10 mg + Placebo | PF-04171327 25 mg + Placebo | Prednisone 5 mg + Placebo | Placebo
Number analyzed (Participants) | 21 | 22 | 21 | 22
10^3 cells per microliter
  Baseline: number analyzed (Participants) | 21 | 22 | 20 | 22
  Baseline | 0.19 (0.115) | 0.19 (0.128) | 0.20 (0.094) | 0.15 (0.077)
  Change at Day 1: 1 hour: number analyzed (Participants) | 21 | 20 | 20 | 22
  Change at Day 1: 1 hour | -0.02 (0.069) | -0.02 (0.060) | -0.02 (0.034) | -0.00 (0.050)
  Change at Day 1: 2 hour: number analyzed (Participants) | 21 | 19 | 19 | 22
  Change at Day 1: 2 hour | -0.01 (0.039) | -0.01 (0.042) | -0.03 (0.038) | -0.00 (0.057)
  Change at Day 1: 3 hour: number analyzed (Participants) | 20 | 19 | 20 | 22
  Change at Day 1: 3 hour | -0.01 (0.039) | -0.01 (0.060) | -0.03 (0.039) | -0.00 (0.057)
  Change at Day 1: 4 hour: number analyzed (Participants) | 21 | 20 | 18 | 22
  Change at Day 1: 4 hour | -0.01 (0.072) | -0.03 (0.079) | -0.04 (0.043) | -0.01 (0.048)
  Change at Day 7: 0 hour: number analyzed (Participants) | 20 | 21 | 20 | 21
  Change at Day 7: 0 hour | -0.03 (0.081) | -0.04 (0.101) | -0.02 (0.055) | 0.00 (0.072)
  Change at Day 7: 1 hour: number analyzed (Participants) | 19 | 20 | 18 | 20
  Change at Day 7: 1 hour | -0.02 (0.050) | -0.03 (0.146) | -0.02 (0.056) | -0.01 (0.081)
  Change at Day 7: 2 hour: number analyzed (Participants) | 19 | 21 | 19 | 21
  Change at Day 7: 2 hour | -0.03 (0.059) | -0.07 (0.121) | -0.04 (0.078) | 0.01 (0.077)
  Change at Day 7: 3 hour: number analyzed (Participants) | 19 | 21 | 19 | 21
  Change at Day 7: 3 hour | -0.04 (0.063) | -0.08 (0.114) | -0.07 (0.087) | 0.00 (0.085)
  Change at Day 7: 4 hour: number analyzed (Participants) | 19 | 20 | 19 | 20
  Change at Day 7: 4 hour | -0.04 (0.070) | -0.06 (0.098) | -0.09 (0.091) | 0.00 (0.080)
  Change at Day 14: 0 hour: number analyzed (Participants) | 17 | 20 | 17 | 19
  Change at Day 14: 0 hour | -0.03 (0.048) | -0.05 (0.167) | -0.02 (0.073) | 0.01 (0.085)
  Change at Day 14: 1 hour: number analyzed (Participants) | 17 | 20 | 19 | 17
  Change at Day 14: 1 hour | -0.04 (0.052) | -0.05 (0.163) | -0.03 (0.076) | -0.01 (0.079)
  Change at Day 14: 2 hour: number analyzed (Participants) | 17 | 20 | 19 | 17
  Change at Day 14: 2 hour | -0.05 (0.063) | -0.07 (0.139) | -0.05 (0.074) | 0.01 (0.092)
  Change at Day 14: 3 hour: number analyzed (Participants) | 17 | 20 | 18 | 16
  Change at Day 14: 3 hour | -0.05 (0.063) | -0.07 (0.139) | -0.09 (0.091) | 0.01 (0.098)
  Change at Day 14: 4 hour: number analyzed (Participants) | 17 | 20 | 18 | 20
  Change at Day 14: 4 hour | -0.05 (0.065) | -0.07 (0.157) | -0.11 (0.096) | -0.01 (0.076)

25. Secondary Outcome: Change From Baseline in Osteocalcin Level at Day 1, 7 and 14
Time Frame: Baseline; 1, 2, 3 and 4 hours post-dose on Day 1; 0, 1, 2, 3 and 4 hours post-dose on Day 7 and 14
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04171327 10 mg + Placebo | PF-04171327 25 mg + Placebo | Prednisone 5 mg + Placebo | Placebo
Number analyzed (Participants) | 21 | 22 | 21 | 22
ng/mL
  Baseline: number analyzed (Participants) | 20 | 22 | 20 | 21
  Baseline | 21.76 (13.031) | 17.52 (9.803) | 29.36 (46.812) | 15.29 (7.156)
  Change at Day 1: 1 hour: number analyzed (Participants) | 20 | 22 | 20 | 21
  Change at Day 1: 1 hour | -1.78 (2.012) | -1.45 (3.164) | -1.94 (2.897) | -0.50 (6.877)
  Change at Day 1: 2 hour: number analyzed (Participants) | 20 | 22 | 20 | 21
  Change at Day 1: 2 hour | -2.22 (2.344) | -2.07 (3.110) | -1.19 (4.445) | -0.73 (3.662)
  Change at Day 1: 3 hour: number analyzed (Participants) | 20 | 22 | 20 | 21
  Change at Day 1: 3 hour | -2.67 (3.063) | -1.07 (2.003) | -1.35 (3.355) | -1.30 (4.150)
  Change at Day 1: 4 hour: number analyzed (Participants) | 20 | 22 | 20 | 21
  Change at Day 1: 4 hour | -3.15 (2.964) | -1.77 (1.849) | -3.10 (5.281) | -0.93 (3.006)
  Change at Day 7: 0 hour: number analyzed (Participants) | 18 | 21 | 19 | 21
  Change at Day 7: 0 hour | -5.26 (5.312) | -3.82 (5.308) | -3.08 (3.995) | 0.69 (3.024)
  Change at Day 7: 1 hour: number analyzed (Participants) | 18 | 21 | 19 | 20
  Change at Day 7: 1 hour | -5.88 (4.719) | -4.42 (7.438) | -0.66 (6.633) | -0.37 (2.976)
  Change at Day 7: 2 hour: number analyzed (Participants) | 18 | 21 | 19 | 20
  Change at Day 7: 2 hour | -5.71 (4.842) | -4.22 (4.765) | -2.74 (5.384) | -0.52 (3.901)
  Change at Day 7: 3 hour: number analyzed (Participants) | 18 | 21 | 19 | 20
  Change at Day 7: 3 hour | -5.77 (7.349) | -3.68 (5.324) | -2.83 (5.194) | -0.33 (4.304)
  Change at Day 7: 4 hour: number analyzed (Participants) | 18 | 21 | 19 | 20
  Change at Day 7: 4 hour | -5.78 (6.145) | -3.87 (5.488) | -2.48 (6.523) | -1.05 (4.206)
  Change at Day 14: 0 hour: number analyzed (Participants) | 18 | 21 | 19 | 19
  Change at Day 14: 0 hour | -6.01 (6.184) | -4.56 (6.155) | -3.04 (6.087) | 0.63 (2.175)
  Change at Day 14: 1 hour: number analyzed (Participants) | 17 | 21 | 19 | 19
  Change at Day 14: 1 hour | -6.28 (6.197) | -4.90 (5.666) | -2.66 (5.289) | -0.25 (2.588)
  Change at Day 14: 2 hour: number analyzed (Participants) | 17 | 21 | 19 | 19
  Change at Day 14: 2 hour | -5.80 (5.833) | -5.11 (6.341) | -4.21 (5.936) | -0.35 (3.507)
  Change at Day 14: 3 hour: number analyzed (Participants) | 17 | 21 | 19 | 19
  Change at Day 14: 3 hour | -6.42 (6.142) | -5.74 (6.195) | -5.88 (10.958) | 0.56 (4.890)
  Change at Day 14: 4 hour: number analyzed (Participants) | 17 | 21 | 18 | 19
  Change at Day 14: 4 hour | -7.45 (7.144) | -5.40 (6.536) | -4.19 (4.398) | -0.41 (4.828)

26. Secondary Outcome: Change From Baseline in Plasma Cortisol Level at Day 1, 7 and 14
Time Frame: Baseline; 1, 2, 3 and 4 hours post-dose on Day 1; 0, 1, 2, 3 and 4 hours post-dose on Day 7 and 14
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04171327 10 mg + Placebo | PF-04171327 25 mg + Placebo | Prednisone 5 mg + Placebo | Placebo
Number analyzed (Participants) | 21 | 22 | 21 | 22
ng/mL
  Baseline: number analyzed (Participants) | 21 | 22 | 21 | 21
  Baseline | 106.85 (27.404) | 110.50 (48.340) | 106.38 (41.396) | 105.14 (56.721)
  Change at Day 1: 1 hour: number analyzed (Participants) | 21 | 22 | 21 | 21
  Change at Day 1: 1 hour | -26.40 (26.238) | -30.94 (26.083) | -13.81 (28.559) | -27.71 (21.432)
  Change at Day 1: 2 hour: number analyzed (Participants) | 21 | 22 | 20 | 21
  Change at Day 1: 2 hour | -29.12 (36.305) | -37.17 (40.260) | -22.81 (36.158) | -32.92 (29.781)
  Change at Day 1: 3 hour: number analyzed (Participants) | 21 | 22 | 21 | 21
  Change at Day 1: 3 hour | -20.05 (42.714) | -24.19 (48.793) | -14.95 (41.651) | -21.80 (39.042)
  Change at Day 1: 4 hour: number analyzed (Participants) | 21 | 22 | 21 | 21
  Change at Day 1: 4 hour | -16.47 (35.633) | -21.05 (55.572) | -21.49 (32.521) | -9.16 (50.832)
  Change at Day 7: 0 hour: number analyzed (Participants) | 19 | 21 | 20 | 21
  Change at Day 7: 0 hour | -92.06 (32.334) | -103.76 (49.618) | 6.72 (24.388) | 7.20 (58.163)
  Change at Day 7: 1 hour: number analyzed (Participants) | 19 | 21 | 20 | 20
  Change at Day 7: 1 hour | -93.92 (30.165) | -104.69 (50.229) | -51.94 (32.569) | -25.39 (44.117)
  Change at Day 7: 2 hour: number analyzed (Participants) | 19 | 21 | 20 | 20
  Change at Day 7: 2 hour | -93.69 (30.420) | -104.96 (50.522) | -66.70 (33.932) | -35.19 (44.417)
  Change at Day 7: 3 hour: number analyzed (Participants) | 19 | 21 | 20 | 20
  Change at Day 7: 3 hour | -94.81 (31.049) | -105.01 (49.683) | -77.36 (33.208) | -26.69 (36.852)
  Change at Day 7: 4 hour: number analyzed (Participants) | 19 | 21 | 20 | 20
  Change at Day 7: 4 hour | -98.82 (26.955) | -104.69 (49.771) | -83.46 (34.019) | -20.38 (43.739)
  Change at Day 14: 0 hour: number analyzed (Participants) | 19 | 21 | 20 | 19
  Change at Day 14: 0 hour | -92.02 (37.108) | -104.86 (50.721) | -14.46 (29.806) | 3.49 (48.156)
  Change at Day 14: 1 hour: number analyzed (Participants) | 18 | 21 | 20 | 19
  Change at Day 14: 1 hour | -98.93 (29.046) | -105.41 (51.193) | -55.14 (39.771) | -25.38 (17.075)
  Change at Day 14: 2 hour: number analyzed (Participants) | 18 | 21 | 20 | 19
  Change at Day 14: 2 hour | -101.65 (27.335) | -105.70 (51.242) | -70.60 (33.658) | -33.54 (30.064)
  Change at Day 14: 3 hour: number analyzed (Participants) | 18 | 21 | 20 | 19
  Change at Day 14: 3 hour | -101.78 (27.765) | -105.29 (51.583) | -81.66 (35.573) | -23.01 (38.787)
  Change at Day 14: 4 hour: number analyzed (Participants) | 18 | 21 | 19 | 19
  Change at Day 14: 4 hour | -102.85 (27.210) | -105.25 (51.263) | -86.27 (37.588) | -24.87 (38.497)

27. Secondary Outcome: Change From Baseline in Ratio of Urinary N-terminal Telopeptide of Type 1 Collagen (uNTX-I) Level to Urinary Creatinine (uCr) Level at Day 7 and 14
Description: Unit of ratio of urinary N-terminal telopeptide of type 1 collagen (uNTX-I) level to urinary creatinine (uCr) level was nanomoles bone collagen equivalents (nmol bce) per millimole creatinine (mmol cr).
Time Frame: Baseline, Day 7 and 14
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: nmol BCE/mmol cr
Arm/Group | PF-04171327 10 mg + Placebo | PF-04171327 25 mg + Placebo | Prednisone 5 mg + Placebo | Placebo
Number analyzed (Participants) | 21 | 22 | 21 | 22
nmol BCE/mmol cr
  Baseline: number analyzed (Participants) | 18 | 21 | 20 | 19
  Baseline | 63.56 (28.239) | 62.00 (26.946) | 77.75 (51.582) | 79.63 (51.794)
  Change at Day 7: number analyzed (Participants) | 16 | 20 | 19 | 19
  Change at Day 7 | 7.94 (16.482) | 16.40 (23.922) | -3.58 (29.632) | -13.42 (31.783)
  Change at Day 14: number analyzed (Participants) | 14 | 20 | 19 | 16
  Change at Day 14 | 11.79 (29.100) | 18.15 (19.626) | -3.84 (33.997) | -9.44 (33.369)

28. Secondary Outcome: Change From Baseline in Adiponectin Level at Day 7 and 14
Time Frame: Baseline, Day 7 and 14
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04171327 10 mg + Placebo | PF-04171327 25 mg + Placebo | Prednisone 5 mg + Placebo | Placebo
Number analyzed (Participants) | 21 | 22 | 21 | 22
ng/mL
  Baseline: number analyzed (Participants) | 21 | 22 | 21 | 21
  Baseline | 7251.43 (3651.564) | 8349.09 (3105.632) | 7732.38 (3428.231) | 10080.95 (5136.660)
  Change at Day 7: number analyzed (Participants) | 19 | 21 | 20 | 21
  Change at Day 7 | -434.21 (3895.367) | 1664.76 (1651.925) | -12.00 (1274.931) | -430.95 (3049.383)
  Change at Day 14: number analyzed (Participants) | 19 | 21 | 20 | 19
  Change at Day 14 | 1023.16 (2203.248) | 2692.86 (2409.083) | 438.50 (951.189) | 193.16 (1965.254)

ADVERSE EVENTS:
Arm/Group | PF-04171327 10 mg + Placebo | PF-04171327 25 mg + Placebo | Prednisone 5 mg + Placebo | Placebo
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/22 | 0/21 | 0/22
Other Adverse Events (participants affected / at risk) | 8/21 | 3/22 | 4/21 | 12/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | PF-04171327 10 mg + Placebo (N=21) | PF-04171327 25 mg + Placebo (N=22) | Prednisone 5 mg + Placebo (N=21) | Placebo (N=22)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Adrenal cyst (Endocrine disorders) | 0 | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 1
Face oedema (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 0 | 0
Irritability (General disorders) | 1 | 0 | 0 | 1
Oedema peripheral (General disorders) | 1 | 1 | 0 | 1
Thirst (General disorders) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Herpes virus infection (Infections and infestations) | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 2 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Blood creatine increased (Investigations) | 0 | 1 | 0 | 0
Blood urea increased (Investigations) | 0 | 1 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 2
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 2 | 4
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0/14 | 1/12 | 0/15 | 0/20 — This event was gender specific.
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Skin lesion (Vascular disorders) | 0 | 0 | 0 | 1
Pallor (Vascular disorders) | 0 | 0 | 0 | 1
Raynaud's phenomenon (Vascular disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.